# I5Q-MC-CGAH (a) Clinical Protocol

A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients with Episodic Migraine – the EVOLVE-2 Study

NCT02614196

Approval Date: 22-Jan-2016

# Protocol I5Q-MC-CGAH(a) A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients with Episodic Migraine – the EVOLVE-2 Study

#### **Confidential Information**

The information contained in this document is confidential and is intended for the use of clinical investigators. It is the property of Eli Lilly and Company or its subsidiaries and should not be copied by or distributed to persons not involved in the clinical investigation of LY2951742, unless such persons are bound by a confidentiality agreement with Eli Lilly and Company or its subsidiaries.

Note to Regulatory Authorities: this document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

#### LY2951742

Study CGAH is a Phase 3, multisite, randomized, double-blind, placebo-controlled, 6-month study to compare the efficacy and safety of two doses of LY2951742 with placebo in preventing migraine headaches in patients with episodic migraine (with or without aura).

Eli Lilly and Company Indianapolis, Indiana USA 46285

Protocol Electronically Signed and Approved by Lilly: 23 September 2015
Protocol Amendment (a) Electronically Signed and Approved by Lilly on approval date provided below.

Approval Date: 22-Jan-2016 GMT

# **Table of Contents**

| Section | Page |
|-------------------------------------------------------|------|
| 1. Protocol Synopsis | 8 |
| 2. Introduction | 11 |
| 2.1. Background | 11 |
| 2.2. Study Rationale | 11 |
| 3. Objectives and Endpoints | 13 |
| 4. Study Design. | 19 |
| 4.1. Overview of Study Design | |
| 4.2. End of Trial Definition | 21 |
| 4.3. Scientific Rationale for Study Design | 21 |
| 4.4. Justification for Dose | 21 |
| 4.5. Benefit/Risk Assessment | 21 |
| 5. Study Population | 22 |
| 5.1. Inclusion Criteria | 22 |
| 5.2. Exclusion Criteria | 23 |
| 5.3. Screen Failures | 26 |
| 5.4. Lifestyle and/or Dietary Requirements | 26 |
| 6. Treatment | 27 |
| 6.1. Treatments Administered | 27 |
| 6.1.1. Medical Devices | 27 |
| 6.2. Method of Treatment Assignment | 27 |
| 6.2.1. Selection and Timing of Doses | 27 |
| 6.3. Blinding | 27 |
| 6.4. Packaging and Labelling | |
| 6.5. Preparation/Handling/Storage. | |
| 6.6. Dose Modification | |
| 6.6.1. Special Treatment Considerations | |
| 6.7. Treatment Compliance | |
| 6.8. Concomitant Therapy | |
| 6.9. Treatment after Study Completion | |
| 6.9.1. Study Extensions. | |
| 6.9.2. Continued Access | |
| 7. Discontinuation Criteria | |
| 7.1. Discontinuation from Study Treatment | |
| 7.1.1. Permanent Discontinuation from Study Treatment | 31 |

| 7.1.2. | Temporary Discontinuation from Study Treatment | 31 |
|------------------|----------------------------------------------------|----|
| 7.1.3. | Discontinuation of Inadvertently Enrolled Patients | 31 |
| 7.1.4. | Permanent Discontinuation from the Study | 32 |
| 7.1.5. | Patients Lost to Follow-Up | 32 |
| 8. Study | y Assessments and Procedures | 33 |
| 8.1. Et | fficacy Assessments | 33 |
| 8.1.1. | Primary Efficacy Assessments | 33 |
| 8.1.2. | Secondary Efficacy Assessments | 33 |
| 8.1.2 | .1. Patient Global Impression of Severity | 33 |
| 8.1.2 | .2. Patient Global Impression of Improvement | 33 |
| 8.1.3. | rr -r | |
| 8.2. A | dverse Events | |
| 8.2.1. | Serious Adverse Events | 34 |
| 8.2.1 | .1. Suspected Unexpected Serious Adverse Reactions | 35 |
| 8.2.1 | | |
| 0.00 | Questionnaire | |
| 8.2.2. | Complaint Handling | |
| | reatment of Overdose | |
| | nfety Assessments | |
| 8.4.1.<br>8.4.2. | Electrocardiograms | |
| 8.4.2.<br>8.4.3. | Vital Signs | |
| 8.4.4. | Laboratory Tests Other Tests | |
| 8.4.5. | Safety Monitoring | |
| | narmacokinetics | |
| | narmacodynamics | |
| | larmacodynamics | 56 |
| 8.8. Bi | iomarkers | 39 |
| 8.8.1. | Samples for Immunogenicity Research. | |
| | ealth Economics | |
| | stical Considerations and Data Analysis | |
| | etermination of Sample Size | |
| | eneral Statistical Considerations | |
| | reatment Group Comparability | |
| 9.3.1. | Patient Disposition | |
| 9.3.2. | Patient Characteristics | |
| 9.3.3. | Concomitant Therapy | |
| 9.3.4. | Treatment Compliance | |

| <b>I5Q-MC-CGAH</b> | (a) | Clinical | Protoco |
|--------------------|-----|----------|---------|
|--------------------|-----|----------|---------|

| 9.3.5. | Electronic Patient-reported Outcome Diary Compliance | 43 |
|---|---|---|
| 9.4. Prin | nary and Secondary Analyses | 43 |
| 9.4.1. | Primary Analyses | 43 |
| 9.4.2. | Key Secondary Analyses | 44 |
| 9.4.3. | Other Secondary and Tertiary Efficacy Analyses | 45 |
| 9.5. Safe | ety Analyses | 46 |
| 9.5.1. | Categorical Safety Variables | 46 |
| 9.5.2. | Adverse Events | 46 |
| 9.5.3. | Suicide-Related Thoughts and Behaviors | 47 |
| 9.5.4. | Vital Signs and Weight | 47 |
| 9.5.5. | Electrocardiogram Intervals and Heart Rate | 47 |
| 9.5.6. | Laboratory Tests | 48 |
| CCI | | |
| | er Analyses | 48 |
| 9.7.1. | Health Economics | 48 |
| 9.7.2. | Subgroup Analyses | 48 |
| 9.8. Inte | rim Analyses | |
| 10. Study ( | Governance Considerations | 51 |
| • | ulatory and Ethical Considerations, Including the Informed | |
| _ | sent Process | 51 |
| 10.1.1. | Informed Consent | 51 |
| 10.1.2. | Ethical Review | 51 |
| 10.1.3. | Regulatory Considerations | 51 |
| 10.1.4. | Investigator Information | 52 |
| 10.1.5. | Protocol Signatures | 52 |
| 10.1.6. | Final Report Signature | 52 |
| 10.2. Data | a Quality Assurance | 52 |
| 10.2.1. | Data Capture System | 53 |
| 10.3. Stud | dy and Site Closure | |
| 10.3.1. | Discontinuation of Study Sites | |
| 10.3.2. | Discontinuation of the Study | |
| | nces | |

### **List of Tables**

| Table | | Page |
|---|---|---|
| Table CGAH.1. | Objectives and Endpoints | 13 |
| Table CGAH.2. | Migraine and Headache Endpoint Definitions | 18 |
| Table CGAH.3. | Treatments Allowed and Treatments Not Allowed as Concomitant Therapy | 29 |
| Table CGAH.4. | Definition of Subgroup Variables | 49 |

# **List of Figures**

| Figure | Page |
|---|---|
| Figure CGAH.1. Illustration of study design for Clinical Protocol I5Q-MC-CGAH | 19 |

# **List of Appendices**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Abbreviations and Definitions | 57 |
| Appendix 2. | Schedule of Activities | 58 |
| Appendix 3. | Clinical Laboratory Tests | 63 |
| Appendix 4. | Hepatic Monitoring Tests for Treatment-Emergent Abnormality | 65 |
| Appendix 5. | Protocol Amendment I5Q-MC-CGAH(a) Summary: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients with Episodic Migraine – the EVOLVE-2 Study | 66 |

# 1. Protocol Synopsis

#### Title of Study:

A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients with Episodic Migraine – the EVOLVE-2 Study.

#### Rationale:

Study I5Q-MC-CGAH (CGAH; EVOLVE-2) is intended to assess the efficacy and safety of two doses of LY2951742 in the prevention of migraine headache compared with placebo in patients suffering from episodic migraine. Episodic migraine is defined as 4 to 14 migraine headache days (with or without aura) per month.

#### **Objective(s)/Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary To test the hypothesis that at least 1 dose of LY2951742 (120 or 240 mg/month) is superior to placebo in the prevention of migraine headache in patients with episodic migraine. | The overall mean change from baseline in the number of monthly migraine headache days during the 6-month double-blind treatment phase |
| Key Secondary Objectives If LY2951742 (120 or 240 mg/month) is statistically significantly superior to placebo on the primary objective, the following key secondary objectives will be tested with adjustment for multiplicity (only the key secondary objectives are listed below): | The specific methodology (including testing order, relationship and type I error allocation and propagation) for the tests of the following key secondary endpoints will be specified in the statistical analysis plan: |
| To compare LY2951742 with placebo with respect to 50% response rate | The proportion of patients with reduction from baseline ≥50% in monthly migraine headache days during the 6-month double-blind treatment phase |
| To compare LY2951742 with placebo with respect to 75% response rate | The proportion of patients with reduction from baseline ≥75% in monthly migraine headache days during the 6-month double-blind treatment phase |
| To compare LY2951742 with placebo with respect to 100% response rate | The proportion of patients with a 100% reduction<br>from baseline in monthly migraine headache<br>days during the 6-month double-blind treatment<br>phase |

| Objectives | Endpoints |
|---|---|
| To compare LY2951742 with placebo with respect to change in functioning | The mean change from baseline in the Role<br>Function-Restrictive domain score of the<br>Migraine-Specific Quality of Life Questionnaire<br>version 2.1 (MSQ v2.1) (average of Months 4, 5, and 6) |
| To compare LY2951742 with placebo with respect<br>to change in use of acute (abortive) migraine<br>treatment | The overall mean change from baseline in the<br>number of monthly migraine headache days<br>requiring medication for the acute treatment of<br>migraine or headache during the 6-month double-<br>blind treatment phase |
| To compare LY2951742 with placebo with respect<br>to change in global severity of the migraine<br>condition | • The mean change from baseline in the Patient<br>Global Impression of Severity (PGI-S) score<br>(average of Months 4, 5, and 6) |

#### **Summary of Study Design:**

A multisite, randomized, double-blind, parallel, placebo-controlled trial with 4 study periods in patients who meet International Classification of Headache Disorders (ICHD) criteria for a diagnosis of migraine as confirmed during a prospective baseline period that demonstrates episodic frequency (4 to 14 migraine headache days per month).

#### **Treatment Arms and Duration:**

Three treatment arms: LY2951742 (120 mg/month with a 240 mg loading dose at the first injection [administered as 2 injections of 120 mg at Visit 3]), LY2951742 (240 mg/month, administered as 2 injections of 120 mg), and placebo. Following a prospective baseline (30-40 days) period, eligible patients will be randomized in a 2:1:1 ratio to receive placebo, 120 mg/month of LY2951742, or 240 mg/month of LY2951742, respectively, and will begin a 6-month treatment phase. This phase will be followed by a 4-month, post-treatment phase during which patients will no longer receive any study medication.

#### **Number of Patients:**

The study will screen an estimated 1557 potential study participants to ensure randomization of approximately 825 patients with episodic migraine.

#### **Statistical Analysis:**

Unless otherwise specified, analyses will be conducted on an intent-to-treat (ITT) population, which include all patients who are randomized and receive at least one dose of investigational product. Patients in the ITT population will be analyzed according to the treatment group to which they are randomized. When mean change from baseline is assessed, the patient will be included in the analysis only if the patient has a baseline and postbaseline measurement.

The primary analysis will evaluate the efficacy of two doses of LY2951742 compared with placebo on the overall mean change from baseline in the number of monthly migraine headache days during the 6-month double-blind treatment phase. Migraine headache day will be defined to include both migraine and probable migraine days. The

primary analysis will be performed using a restricted maximum likelihood based mixed models repeated measures (MMRM) technique. The analysis will include the fixed categorical effects of treatment, region, month, and treatment-by-month interaction, as well as the continuous fixed covariates of baseline number of migraine headache days and baseline number of migraine headache days-by-visit interaction.

## 2. Introduction

# 2.1. Background

Migraine is a chronic, debilitating condition found to be one of the top 10 causes of disability expressed as years lived with disability globally (Vos et al. 2012). However, one study estimates that only a small fraction of patients receive preventive treatment, although more than 25% of migraineurs are in need of preventive therapy (Rizzoli 2014). Despite the availability of preventive medications for migraine, significant needs remain for new treatment options with improved efficacy and tolerability.

Calcitonin gene-related peptide (CGRP), a 37-amino acid neuropeptide, is widely expressed throughout the central and peripheral nervous system and acts as a local facilitator of inflammatory processes. CGRP is implicated in the pathophysiology of migraine and is hypothesized to be involved in the release of inflammatory mediators and the transmission of nociceptive (pain) information from intracranial blood vessels to the nervous system (Villalón and Olesen 2009). In migraineurs, serum concentrations of CGRP are significantly elevated during migraine attacks (Goadsby et al. 1990; Goadsby and Edvinsson 1993), and infusion of CGRP to individuals with a history of migraine can trigger migraine attacks (Lassen et al. 1998; Lassen et al. 2002). The neutralization of CGRP with antibodies has been shown to modulate neurogenic inflammation; thus, these antibodies may represent a promising pharmacologic approach for the prevention of migraine (Investigator's Brochure [IB], Section 3.1).

LY2951742 is a humanized monoclonal antibody that potently and selectively binds to CGRP, preventing CGRP-mediated biological effects (IB, Section 3.1). To date, more than 450 clinical trial participants have been exposed to LY2951742 at single doses ranging from 1 to 600 mg and multiple doses up to 300 mg in 5 clinical trials of LY2951742. In studies of patients with migraine (Studies I5Q-MC-ART1 [ART-01] and I5Q-MC-CGAB [CGAB]), efficacy data have demonstrated that LY2951742 had significantly greater mean reductions than placebo in migraine headache days and other efficacy parameters. Across clinical studies of LY2951742, assessment of adverse events (AEs) indicates that LY2951742 has been well tolerated in both healthy subjects and in patients with episodic migraine. The AEs generally have been mild to moderate in severity. In two studies of patients with migraine, the most frequently reported adverse events (AEs) included injection-site pain, upper respiratory tract infection, abdominal pain, dizziness, injection-site erythema, rash, hypertension, and nasopharyngitis. Analyses of laboratory values and cardiovascular monitoring of the clinical studies have shown no other clinically important changes in tested parameters.

# 2.2. Study Rationale

Study I5Q-MC-CGAH (EVOLVE-2) will enable a more comprehensive clinical assessment of LY2951742 in a patient population for which the drug already has shown preliminary evidence of efficacy and safety. This study, along with a study of identical design in patients with episodic migraine, is intended to provide pivotal efficacy data to support a registration program in patients with migraines. EVOLVE-2 will include 6 months on LY2951742 or placebo

followed by 4 months of post-treatment observation to deepen understanding of the effects of a CGRP antibody in preventing migraines.

# 3. Objectives and Endpoints

Table CGAH.1 shows the key objectives and endpoints of the study. Table CGAH.2 provides definitions for the terms referenced below.

Table CGAH.1. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary To test the hypothesis that at least 1 dose of LY2951742 (120 or 240 mg/month) is superior to placebo in the prevention of migraine headache in patients with episodic migraine. | The overall mean change from baseline in the number of monthly migraine headache days during the 6-month double-blind treatment phase |
| Key Secondary Objectives If LY2951742 (120 or 240 mg/month) is statistically significantly superior to placebo on the primary objective, the following key secondary objectives will be tested with adjustment for multiplicity: | The specific methodology (including testing order, relationship and type I error allocation and propagation) for the tests of the following key secondary endpoints will be specified in the statistical analysis plan: |
| To compare LY2951742 with placebo with respect to 50% response rate | • The proportion of patients with reduction from baseline ≥50% in monthly migraine headache days during the 6-month double-blind treatment phase |
| To compare LY2951742 with placebo with respect<br>to 75% response rate | • The proportion of patients with reduction from baseline ≥75% in monthly migraine headache days during the 6-month double-blind treatment phase |
| To compare LY2951742 with placebo with respect<br>to 100% response rate | The proportion of patients with a 100% reduction<br>from baseline in monthly migraine headache days<br>during the 6-month double-blind treatment phase |
| To compare LY2951742 with placebo with respect to change in functioning | • The mean change from baseline in the Role Function-Restrictive domain score of the Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ v2.1) (average of Months 4, 5, and 6) |

Table CGAH.1. Objectives and Endpoints (continued)

| Objectives (cont.) | | Endpoints (cont.) | |
|---|---|---|---|
| Ke | y Secondary Objectives (cont.) | | |
| • | To compare LY2951742 with placebo with respect to change in use of acute (abortive) migraine treatment | • | The overall mean change from baseline in the number of monthly migraine headache days requiring medication for the acute treatment of migraine or headache during the 6-month doubleblind treatment phase |
| • | To compare LY2951742 with placebo with respect to change in global severity of migraine condition | • | The mean change from baseline in the Patient Global Impression of Severity (PGI-S) score (average of Months 4, 5, and 6) |
| Ot | her Secondary Objectives | | |
| • | To compare LY2951742 with placebo with respect to change in headache days | • | The overall mean change from baseline in the number of monthly headache days during the 6-month double-blind treatment phase |
| • | To compare LY2951742 with placebo with respect to change in moderate to severe headache days | • | The overall mean change from baseline in the number of monthly moderate to severe headache days during the 6-month double-blind treatment phase |
| • | To compare LY2951742 with placebo with respect to a 30% response rate | • | The proportion of patients with reduction from baseline $\geq 30\%$ in monthly migraine headache days during the 6-month double-blind treatment phase |
| • | To compare LY2951742 with placebo with respect to distribution of response rates | • | Cumulative distribution of monthly migraine headache day response rates during the 6-month double-blind treatment phase |
| • | To compare LY2951742 with placebo with respect to time to 50% response | • | Time to first occurrence of a ≥50% reduction from baseline in the number of monthly migraine headache days (Kaplan-Meier analysis) |
| • | To compare LY2951742 with placebo with respect to onset of effect | • | The initial month at which statistical separation in mean change from baseline in the number of monthly migraine headache days is demonstrated and maintained at all subsequent months through Month 6 |
| • | To compare LY2951742 with placebo with respect to onset of 50% sustained response | • | The initial month at which statistical separation in the proportion of patients meeting at least a 50% reduction in monthly migraine headache days that is maintained at all subsequent months through Month 6 |

Table CGAH.1. Objectives and Endpoints (continued)

| Objectives (cont.) Endpoints (cont.) | |
|---|---|
| Other Secondary Objectives (cont.) To compare LY2951742 with placebo with respect to maintenance of 50% response | The proportion of patients who maintain 50% response criteria for at least 3 consecutive months to the end of the double-blind treatment phase and the proportion of patients who maintain 50% response criteria for 6 consecutive months during double-blind treatment |
| <ul> <li>To compare LY2951742 with placebo with respect to changes in other efficacy parameters, specifically: <ul> <li>International Classification of Headache Disorders (ICHD) migraine headache days</li> <li>migraine attacks</li> <li>migraine headache hours</li> <li>headache hours</li> <li>severity of remaining migraines</li> </ul> </li> </ul> | Overall mean change from baseline (during the 6-month double-blind treatment phase) on the following monthly measures: International Classification of Headache Disorders (ICHD) migraine headache days migraine attacks migraine headache hours headache hours severity of remaining migraines |
| To compare LY2951742 with placebo with respect<br>to global assessment of illness | Overall mean Patient Global Impression-<br>Improvement (PGI-I) rating during the 6-month<br>double-blind treatment phase |
| To compare LY2951742 with placebo with respect to changes in disability and quality of life | Mean change from baseline on the following measures: the Migraine Disability Assessment test (MIDAS) total score and individual items at Month 6 the Migraine-Specific Quality of Life Questionnaire, version 2.1 (MSQ v2.1) total score, and Role Function-Preventive and Emotional Function domain scores(average of Months 4, 5, and 6) |
| To compare LY2951742 with placebo with respect<br>to safety and tolerability | Analysis of: treatment-emergent adverse events (TEAEs) discontinuation rates vital signs and weight electrocardiograms (ECGs) laboratory measures other safety parameters, including suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) |

Table CGAH.1. Objectives and Endpoints (continued)

| Objectives (cont.) | Endpoints (cont.) |
|---|---|
| Other Secondary Objectives (cont.) To evaluate LY2951742 with respect to immunogenicity | <ul> <li>Throughout the study:</li> <li>Development and consequences of anti-drug antibodies and neutralizing anti-drug antibodies to LY2951742</li> </ul> |
| To evaluate LY2951742 with respect to<br>pharmacokinetics | Serum concentrations of LY2951742 |
| To evaluate LY2951742 with respect to<br>pharmacodynamics (target engagement) | Plasma concentrations of CGRP |
| To assess changes in efficacy outcomes during<br>Study Period IV as collected by electronic patient-<br>reported outcomes (ePRO) diary data | In Study Period IV: Mean change from baseline in monthly migraine headache days Time to first loss of response among patients who met the 50% response rate criteria at the end of the double-blind treatment phase Time to initiation of treatment with a migraine prevention medication |
| Tertiary Objectives | |
| CCI | |
| To explore the effect of LY2951742 on non-<br>migraine chronic pain | Mean change from baseline in average pain severity<br>of other chronic pain conditions |
| To compare LY2951742 with placebo with respect<br>to categorical changes in quality of life | <ul> <li>Percentages of patients with: <ul> <li>≥50% improvement in MIDAS total score</li> <li>change from baseline in MSQ Role Function-Restrictive domain ≥10.9</li> <li>change from baseline in MSQ Role Function-Preventive domain ≥8.3</li> <li>change from baseline in MSQ Emotional Function domain ≥12.2</li> </ul> </li> </ul> |

Table CGAH.1. Objectives and Endpoints (continued)

| Objectives (cont.) | Endpoints (cont.) |
|---|---|
| Tertiary Objectives (cont.) To compare LY2951742 with placebo with respect to the proportion of migraine headache days requiring medication for the acute treatment of migraine or headache | Change from baseline in the proportion of monthly migraine headache days requiring medication for the acute treatment of migraine or headache |
| To compare LY2951742 with placebo with respect<br>to changes in symptomatology associated with<br>migraine or probable migraine | <ul> <li>Change from baseline in the number of monthly migraine headache days with:</li> <li>nausea and/or vomiting</li> <li>photophobia and phonophobia</li> <li>aura</li> <li>prodromal symptoms other than aura</li> </ul> |

 Table CGAH.2.
 Migraine and Headache Endpoint Definitions

| Diagnosis | Definition/Criteria |
|---|---|
| Migraine headache | A headache, with or without aura, of ≥30 minutes duration with both of the following required features (A and B): A. At least 2 of the following headache characteristics: |
| | Unilateral location |
| | Pulsatile quality |
| | Moderate or severe pain intensity |
| | Aggravation by or causing avoidance of routine physical activity |
| | AND |
| | B. During headache at least one of the following: |
| | Nausea and/or vomiting |
| | Photophobia and phonophobia |
| | (Definition adapted from the Standard International<br>Headache Society [IHS] International Classification of<br>Headache Disorders (ICHD)-3 beta) |
| Probable migraine | A headache missing 1 of the migraine features in the IHS |
| | ICHD-3 beta definition such that one feature in criteria A is missing or one feature in criteria B is missing; that is, meet at least 2 A criteria and none of the B criteria or meet 1 of the A |
| | criteria and at least 1 of the B criteria. |
| Migraine headache day (primary objective) | A calendar day on which a migraine headache or probable migraine headache occurred. |
| Migraine headache attack | Beginning on any day a migraine headache or probable migraine headache is recorded and ends when a migraine-free day occurs. |
| Non-migraine headache | All headaches of at least 30 minutes duration not fulfilling the definition of migraine or probable migraine are classified as non-migraine headaches. |
| Non-migraine headache day | A calendar day on which a non-migraine headache occurred. |
| Headache day | A calendar day on which any type of headache occurs (including migraine headache, probable migraine headache, and non-migraine headache). |

# 4. Study Design

# 4.1. Overview of Study Design

Study CGAH (EVOLVE-2) is a Phase 3, multisite, double-blind, randomized, placebo-controlled, study of LY2951742 in patients suffering from episodic migraine. The study has 4 periods, including a prospective baseline phase to determine patient eligibility.

Figure CGAH.1 illustrates the study design.



<sup>\*</sup>Eligibility period determined between a minimum of 30 days and a maximum of 40 days. Investigators may have up to 5 additional days (beyond the 40 days) if needed to schedule patients' Visit 3 appointment.

Figure CGAH.1. Illustration of study design for Clinical Protocol I5Q-MC-CGAH.

**Study Period I**: The study and potential risks will be explained to the patient at Visit 1. The informed consent form (ICF) must be signed before any study procedures are performed. Patients are required to discontinue all excluded medications or migraine prevention treatments at least 30 days prior to Visit 2. Botulinum toxin A or B in the head or neck area must be discontinued at least 4 months prior to Visit 2.

<sup>&</sup>lt;sup>a</sup>Patients randomized to the 120 mg dose will receive a loading dose of 240 mg at the first injection only (Visit 3). Abbreviations: SP = study period.

The screening visit (Visit 1) will consist of a full clinical assessment, including a comprehensive medical evaluation documenting medical history, and a physical and neurological examination (Appendix 2). Visit 1 will be complete when the last scheduled procedure of the screening assessment is completed.

**Study Period II**: Qualified patients will enter Study Period II (prospective baseline) to determine their eligibility for the study and to establish baseline data for comparison of endpoints during the treatment period. Beginning at Visit 2, patients will log in daily to the electronic patient-reported outcomes (ePRO) system to answer questions about the occurrence of headaches, headache duration, headache features, severity of headache, and use of headache medication. At the end of the prospective baseline period, sites will be notified whether their patients met criteria and are eligible to be randomized at Visit 3.

To avoid biased reporting, patients must not be told the number of migraine headache days on which study qualification is based.

**Study Period III**: At the start of the 6-month double-blind treatment phase (Visit 3), patients meeting all eligibility requirements will be randomized to 1 of 3 treatment groups in a 2:1:1 ratio to receive placebo, 120 mg/month LY2951742, or 240 mg/month LY2951742, respectively.

Patients randomized to the 120 mg dose of LY2951742 will receive an initial loading dose of 240 mg (2 injections of 120 mg each at Visit 3 only). To preserve blinding throughout the study, patients in all treatment groups will receive 2 injections of investigational product at each dosing visit (two placebo injections, two 120-mg LY2951742 injections, or one placebo injection and one 120-mg injection). At Visit 3, if available and where local regulations and Ethical Review Boards allow, patients will also watch a training video designed to address patient expectations with regard to participation in a placebo-controlled trial and the difference between medical treatment and research.

The patient will be considered enrolled in the study when randomization occurs. During this phase, study procedures at dosing visits must always occur prior to the patient receiving their assigned treatment.

Patients will be given injections of investigational product during office visits (Figure CGAH.1). For all treatment groups, subcutaneous injections will be administered once monthly at the dosing visits. At Visit 3 (first dose), patients will be required to remain in the office for observation for 30 minutes post injection. Patients will continue to log in and complete the ePRO diary each day. Patients may continue to take their allowed acute migraine headache medication (with some limitations; see Section 6.8) during the treatment phase.

Patients who complete this phase or discontinue for any reason during Study Period III will be expected to enter post-treatment follow-up (Study Period IV).

**Study Period IV**: During this 4-month phase, sites and patients will remain blinded to patients' treatment assignments. Patients will follow all study procedures during Study Period IV but will not receive LY2951742 or placebo. One month after Visit 12, if clinically warranted due to a worsening of symptoms, patients may start migraine prevention medications at the discretion of

the investigator. The list of allowed preventive medications is provided in Section 6.8. At Visit 14 (Month 10), patients will return to the site for their last study visit and discharge from the study.

### 4.2. End of Trial Definition

End of the trial is the date of the last visit or last scheduled procedure shown in the Schedule of Activities (Appendix 2) for the last patient.

## 4.3. Scientific Rationale for Study Design

The length of the randomized treatment phase is considered sufficient to assess the safety and efficacy of a migraine prevention medication and is consistent with regulatory feedback. A 4-month post-treatment follow-up phase is included to evaluate patient safety during wash-out of LY2951742. This allows for a total of 5 months of observation from the time of last injection of LY2951742. A 5-month post-treatment observation period allows for a wash-out of approximately 5 elimination half-lives of LY2951742 and should decrease LY2951742 serum concentrations by approximately 97% during this time.

#### 4.4. Justification for Dose

Doses of 120 and 240 mg administered once monthly were selected primarily on the basis of clinical efficacy and pharmacokinetic/pharmacodynamic data from the Phase 2 dose-ranging study. Results from the Phase 2 dose-ranging study indicate that 120 mg was statistically significantly superior to placebo at the last 28-day period of the 3-month treatment phase in mean change in migraine headache days, as well as in other measures of efficacy and quality of life. The use of a loading dose for the 120 mg treatment arm, and the inclusion of a 240 mg treatment arm, is based on the finding that a dose higher than 120 mg achieved statistically significant separation from placebo as early as Month 1. The planned doses of 120 mg and 240 mg LY2951742 for Study CGAH also are being evaluated in two other pivotal efficacy studies of LY2951742; one of these studies is in patients with episodic migraine, and one is in patients with chronic migraine.

#### 4.5. Benefit/Risk Assessment

More information about the known and expected benefits, risks, serious adverse events (SAEs) and reasonably anticipated adverse events (AEs) of LY2951742 are to be found in the Investigator's Brochure (IB).

# 5. Study Population

All patients must meet the following selection criteria. Eligibility of patients for study enrollment will be based on the results of a screening medical history, physical examination, neurological examination, clinical laboratory tests, electrocardiograms (ECGs), and migraine history during screening and a prospective baseline period, as described in the Inclusion and Exclusion Criteria sections. The nature of any comorbid conditions present at the time of the physical examination and any pre-existing conditions must be documented. Individuals who do not meet the criteria for participation in this study (screen failure) for specific reasons as outlined may be considered for rescreening once, with approval from Eli Lilly and Company (Lilly) Medical (Section 5.3).

Study participants should be instructed not to donate blood or blood products during the study or for 5 months following last administration of investigational product.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, are not permitted.

#### 5.1. Inclusion Criteria

Patients are eligible to be included in the study only if they meet all of the following criteria at screening:

#### **Patient and Disease Characteristics**

- [1] Patients are 18 to 65 years of age (inclusive) at the time of screening.
- [2] Have a diagnosis of migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.1 or 1.2) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to Visit 1, and migraine onset prior to age 50.
- [3] Prior to Visit 1, have a history of 4 to 14 migraine headache days and at least 2 migraine attacks per month on average within the past 3 months.
- [4] From Visit 2 to Visit 3 (prospective baseline period), have a frequency of 4 to 14 migraine headache days and at least 2 migraine attacks (see definitions, Table CGAH.1). To avoid biased reporting, patients must not be told the number of migraine headache days on which study qualification is based.
- [5] From Visit 2 to Visit 3 (prospective baseline period), must achieve sufficient compliance with ePRO daily headache entries as demonstrated by completion of at least 80% of daily diary entries.

## **Informed Consent and Patient Agreements**

- [6] Are able and willing to give signed informed consent.
- [7] Are reliable and willing to follow study procedures, including all follow-up visits.

- [8] Women of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test.
- [9] All patients, male and female, must agree to use a reliable method of birth control during the study as well as for 5 months after the last dose of investigational product. Acceptable methods of birth control for this study include: oral contraceptives; implantable contraceptives; injectable contraceptives; a contraceptive patch; barrier methods such as diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, or intrauterine devices; a partner with vasectomy. Birth control is not required if the female is infertile due to surgical sterilization (at least 6 weeks after surgical bilateral oophorectomy, hysterectomy, or at least 6 weeks after tubal ligation) confirmed by medical history or menopause. Menopause is defined as spontaneous amenorrhea for at least 12 months not induced by a medical condition, or spontaneous amenorrhea of 6-12 months and a follicle stimulating hormone level >40 mIU/mL.
- [10] Agree not to post any personal medical data related to the study or information related to the study on any website or social media site (for example, Facebook, Twitter, LinkedIn, Google+, etc.) until the entire trial has completed.

#### 5.2. Exclusion Criteria

Patients will be excluded from study enrollment if they meet any of the following criteria at screening:

#### **Prior/Concurrent Clinical Trial Experience**

- [11] Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
- [12] Have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product. If the investigational product's half-life is not known, 6 months should have passed prior to Visit 1.
- [13] Current use or prior exposure to LY2951742 or another CGRP antibody, including those who have previously completed or withdrawn from this study or any other study investigating a CGRP antibody.

#### **Prior/Concomitant Therapy**

[14] Patients who are taking, or are expected to take, therapeutic antibodies during the course of the study (for example, adalimumab, infliximab, trastuzumab, bevacizumab, etc.). Prior use of therapeutic antibodies, other than antibodies to CGRP or its receptor, is allowed if that use was more than 12 months prior to Visit 2.

- [15] Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to LY2951742.
- [16] Are currently receiving medication or other treatments for the prevention of migraine headaches. Patients must have discontinued such treatment at least 30 days prior to Visit 2. Botulinum toxin A and B that has been administered in the head or neck area must be discontinued at least 4 months prior to Visit 2.
- [17] Failure to respond to 3 or more adequately dosed migraine preventive treatments from different classes (that is, maximum tolerated dose for at least 2 months). Failure to respond due to tolerability issues is not considered a treatment failure. Migraine preventive treatments are defined as Level A and Level B in Table 1 of the American Academy of Neurology's Evidence-based Guidelines Update: Pharmacologic Treatment for Episodic Migraine Prevention in Adults (Silberstein et al. 2012) as well as botulinum toxin A or B

#### **Diagnostics Assessments**

- [18] History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.
- [19] History of headache (for example, cluster headache, Medication Overuse Headache) other than migraine or tension type headache as defined by IHS ICHD-3 beta within 3 months prior to randomization.
- [20] Prior to Visit 1, a history of ≥15 headache days (migraine, probable migraine or any other headache) per month on average during the past 3 months or are suspected of suffering from chronic migraine as defined per ICHD-3 beta.
- [21] History of head or neck injury within 6 months prior to Visit 1.
- [22] Patients with a history of traumatic head injury associated with significant change in the quality or frequency of their headaches should be excluded.

#### **Medical Conditions**

- [23] Have ECGs showing abnormalities compatible with acute cardiovascular events and/or serious cardiovascular risk, including but not limited to a corrected QT (QTcB [Bazett's]) interval > 470 msec for women and >450 for men, or have had myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, or deep vein thrombosis/pulmonary embolism within 6 months of screening, or have planned cardiovascular surgery or percutaneous coronary angioplasty, or patients with a lifetime history of stroke.
- [24] Patients with a body mass index  $\geq$ 40 kg/m<sup>2</sup>.

- [25] Any liver tests outside the normal range at Visit 1 that are clinically significant. Alanine aminotransferase (ALT) >2X upper limit of normal (ULN), or total bilirubin (TBL) >1.5X ULN, or alkaline phosphatase (ALP) >2X ULN must be discussed and judged not clinically significant by Lilly Medical prior to enrollment.
- [26] Evidence of significant active or unstable psychiatric disease by medical history, such as bipolar disorder, schizophrenia, personality disorders, or other serious mood or anxiety disorders. Note: Patients with major depressive disorder or generalized anxiety disorder whose disease state is considered stable and expected to remain stable throughout the course of the study, in the opinion of the investigator, may be considered for inclusion if they are not on excluded medications.
- [27] Patients who, in the clinician's judgment, are actively suicidal and therefore deemed to be at significant risk for suicide, or those who have answered "yes" to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the Columbia Suicide Severity Rating Scale (C–SSRS), or answer "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior" portion of the C–SSRS; and the ideation or behavior occurred within the past month.
- [28] Women who are pregnant or nursing.
- [29] Patients who have used opioids or barbiturate containing analgesic >2X per month for the treatment of pain in more than 2 of the past 6 months (opioid administration in an emergency setting may be an exception).
- [30] History of drug or alcohol abuse/dependence within 1 year prior to Visit 1 (excessive or compulsive use as judged by the Investigator), or currently using drugs of abuse (including opioids, barbiturates and marijuana), or any prescribed or over-the-counter medication in a manner that the Investigator considers indicative of abuse/dependence.
- [31] Have a positive urine drug screen for any substances of abuse at Visit 1. Note: A retest is allowed if the urine drug screen is positive for any prescribed substance or if, in the judgment of the investigator, there is an acceptable explanation for the positive result. The results of the retest must be negative at or prior to Visit 2.
- [32] Have a history or presence of any other medical illness including but not limited to any autoimmune disorder, cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, or any clinically significant laboratory abnormality, that in the judgment of the investigator, indicates a medical problem that would preclude study participation.

#### Other Exclusions

- [33] In the opinion of the investigator have other issues which would interfere with compliance with the study requirements and completion of evaluations required for this study.
- [34] Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
- [35] Are Lilly employees.
- [36] Are unwilling or unable to comply with the use of a data collection device.

#### 5.3. Screen Failures

Individuals who do not meet the criteria for participation in this study (screen failure) may be considered for rescreen once, with approval from Lilly Medical for only the criteria shown below. The interval between screening and rescreening must be at least 45 days or longer if required for the specified timeframes in the inclusion/exclusion criteria or concomitant medications requirements. If rescreening is performed, the individual must sign a new ICF and will be assigned a new identification number.

- Inclusion criterion 1. If patients are less than age 18 at time of informed consent, they may be rescreened if they reach age 18 during the study enrollment period.
- Inclusion criterion 8
- Exclusion criterion 12
- Exclusion criterion 14
- Exclusion criterion 16
- Exclusion criterion 28

Patients using a concomitant medication that requires a stable dose for a specific duration prior to Visit 2 may be rescreened if additional time is needed to meet the duration requirement.

In addition, after consultation with and approval by a Lilly Medical representative, a patient may be rescreened if there is an unexpected technical difficulty with the electronic diary capture during the prospective baseline period.

# 5.4. Lifestyle and/or Dietary Requirements

No changes in lifestyle or dietary requirements are required during the study. However, patients must be in a fasting state for collection of laboratory samples at selected visits specified in Appendix 2.

#### 6. Treatment

#### 6.1. Treatments Administered

This study involves a comparison of LY2951742 (120 and 240 mg) administered once monthly with placebo. Sites will administer injections of investigational product (LY2951742 and/or placebo) at 6 office visits during the treatment phase (Appendix 2).

Possible injection sites include the abdomen, thigh, and upper arm. Buttocks may also be used, if needed.

The investigator or his/her designee is responsible for the following:

- maintaining accurate records of investigational product dispensing
- at the end of the study returning all unused medication to Lilly, or its designee, unless the sponsor and sites have agreed all unused medication is to be destroyed by the site, as allowed by local law.

#### 6.1.1. Medical Devices

The manufactured medical devices provided for use in the study are prefilled syringes.

## 6.2. Method of Treatment Assignment

Patients who meet all criteria for enrollment will be randomized to double-blind treatment at Visit 3. Assignment to treatment groups will be determined by a computer-generated random sequence using an interactive web-response system (IWRS). The IWRS will be used to assign double-blind investigational product to each patient. Site personnel will confirm that they have located the correctly assigned package by entering the confirmation number found on the package into the IWRS.

To achieve between-group comparability, the randomization will be stratified by country and baseline migraine frequency (<8 migraine headache days versus  $\ge8$  migraine headache days). To ensure an appropriate balance of low- and high-frequency migraine headache day patients, the sponsor will stop enrollment of low-frequency patients if the number exceeds an estimated 578.

# 6.2.1. Selection and Timing of Doses

This is a fixed-dose study. The actual time of all dose administrations will be recorded in the patient's electronic case report form (eCRF).

# 6.3. Blinding

This is a double-blind study.

To preserve the blinding of the study, a minimum number of Lilly personnel will see the randomization table and treatment assignments before the study is complete.

Emergency unblinding for AEs may be performed through the IWRS. This option may be used ONLY if the patient's well-being requires knowledge of the patient's treatment assignment. All unblinding events are recorded and reported by the IWRS.

If an investigator, site personnel performing assessments, or patient is unblinded, the patient must be discontinued from the study. In cases where there are ethical reasons to have the patient remain in the study, the investigator must obtain specific approval from a Lilly clinical research physician (CRP) or clinical research scientist (CRS) for the patient to continue in the study.

In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a patient's treatment assignment is warranted. Patient safety must always be the first consideration in making such a determination. If an emergency unblinding occurs, Lilly must be notified as soon as possible.

# 6.4. Packaging and Labelling

LY2951742 and matching placebo (excipients only) will be supplied as an injectable solution in 1-mL, single-dose, prefilled, disposable manual syringes with study specific labels. Each syringe of LY2951742 is designed to deliver LY2951742 120 mg. The syringes (and contents) containing either LY2951742 or placebo will be visibly indistinguishable from each other. Syringes will be supplied in cartons, with the appropriate quantity of syringes specific to the planned dispensing schedule of investigational product.

Clinical trial materials will be labeled according to the country's regulatory requirements.

# 6.5. Preparation/Handling/Storage

Investigational product will be shipped (as prefilled syringes) to sites using cold chain transportation. Investigational product must be stable and stored in a refrigerator at 2°C to 8°C (35.6°F to 46.4°F).

Approximately 30 minutes prior to administration, the syringe should be removed from the storage area and allowed to equilibrate at ambient conditions. The drug product should be kept away from direct exposure to bright light (such as sunlight) and hot surfaces until administration.

#### 6.6. Dose Modification

Dose modifications are not permitted in this study.

# 6.6.1. Special Treatment Considerations

During the post-treatment follow-up period, patients will not receive LY2951742 or placebo. One month after Visit 12, if clinically warranted due to a worsening of symptoms, patients may start migraine prevention medications at the discretion of the investigator. The list of allowed preventive medications is provided separately.

# 6.7. Treatment Compliance

Investigators will be required to document the administration of investigational product in the eCRF.

Investigational product must be administered as indicated in the Schedule of Activities (Appendix 2). If the investigator is unable to administer the investigational product in the allowed window, then the situation should be discussed with Lilly to determine if the patient may continue

# 6.8. Concomitant Therapy

Table CGAH.3 contains a list of medications that are, and are not, allowed in this study. Note that acute treatment of migraine headache is allowed throughout the study but with some limitations. Treatments used for the prevention of migraine are not allowed at any time during Study Periods I through III.

# Table CGAH.3. Treatments Allowed and Treatments Not Allowed as Concomitant Therapy

# Medications allowed for the ACUTE treatment of migraine headaches or other pain or injury:

Acetaminophen (paracetamol), NSAIDs; Triptans; Ergotamine and derivatives; Isometheptene mucate, dichloralphenazone and acetaminophen combination (Midrin); or combinations thereof.

The following medications are allowed with restrictions:

- 1. Opioid and barbiturates no more than 3 days/month (SP II, III and IV).
- 2. Single dose of injectable steroids allowed only once during the study, in an emergency setting (SP III and IV).

#### Medications, Procedures or Devices not allowed for any reason/indication:

Acetazolamide

Acupuncture

Anticonvulsants/Antiepileptics

Antipsychotics

Beta-blockers

Botulinum toxin applied to head/neck area

Cannabis / Cannabinoids

Chiropractic procedures, physiotherapy, TENS or other electric devices on head and neck

Corticosteroids for oral use

Flunarizine

Herbals with anti-inflammatory effect (feverfew, willow bark, petasites/butterbur), herbals with sympathomimetic effect (ma huang, ephedra, bitter orange, synephrine) and herbals with catecholamine transmitter reuptake inhibition (St John's Wort)

Monoamine oxidase inhibitors (MAOIs)

Memantine

Serotonin 5HT2a/2c antagonists, e.g.: trazodone, nefazodone

Stimulants (prescription strength), e.g.: methylphenidate, dextroamphetamine, mixed amphetamine salts

Tizanidine

Therapeutic antibodies, e.g.: adalimumab, infliximab, trastuzumab, bevacizumab, etanercept, etc.

Tricyclic antidepressants (TCAs)

Triptans for prophylaxis of menstrual related migraine

Venlafaxine

Verapamil

# Table CGAH.3. Treatments Allowed and Treatments Not Allowed as Concomitant Therapy (continued)

# Restricted medication during SP II-III: Use of the following medications for indications other than migraine prevention is allowed providing the dose is stable 2 months prior to Visit 2 and is expected to remain stable during Visit 2 through 12.

ACE inhibitors

Angiotensin receptor blockers (ARBs)

Benzodiazepines

Bupropion

Calcium-channel blockers (except verapamil and flunarizine)

Clonidine

Guanfacine

Mirtazapine

SSRIs/NRIs/SNRIs (other than venlafaxine)

Use of electric devices (i.e. TENS), physiotherapy, chiropractic procedures on low back and extremities

# Restricted medication during SP II-III: Use of the following medications for indications other than migraine prevention is allowed:

Beta-blockers, ophthalmic

Cyclandelate

Cyproheptadine

Melatonin

#### SP IV (After Visit 12)

One month after Visit 12, if clinically warranted due to a worsening of symptoms, patients may start migraine prevention medications at the discretion of the investigator with the exception of antipsychotics, cannabis and cannabinoids, MAOIs, memantine, serotonin 5HT2a/2c antagonists, and stimulants, which remain excluded.

# 6.9. Treatment after Study Completion

# 6.9.1. Study Extensions

Not applicable.

#### 6.9.2. Continued Access

Investigational product will not be made available to patients after conclusion of the study.

#### 7. Discontinuation Criteria

Patients who discontinue the study or investigational product during the double-blind treatment phase (Study Period III) will proceed immediately to Study Period IV.

# 7.1. Discontinuation from Study Treatment

# 7.1.1. Permanent Discontinuation from Study Treatment

Discontinuation of the investigational product is required in cases of pregnancy.

Discontinuation of the investigational product for abnormal liver tests is required when a patient meets one of the following conditions and the event is at least possibly related to study drug:

- ALT or aspartate aminotransferase (AST) >8X ULN
- ALT or AST >5X ULN for more than 2 weeks
- ALT or AST >3X ULN and TBL >2X ULN or prothrombin time >1.5X ULN
- ALT or AST >3X ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)
- ALP >3X ULN
- ALP >2.5X ULN and TBL >2X ULN
- ALP >2.5X ULN with the appearance of fatigue, nausea, vomiting, right quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)

Discontinuation of investigational product also is required in the following cases, if the event is at least possibly related to study drug:

- Serious allergic reaction to study drug
- Serious injection-site reaction
- Serious event of suicidality or depression
- Serious cerebrovascular event.

Patients who discontinue the investigational product early will have end-of-therapy (early termination) procedures performed as shown in the Schedule of Activities (Appendix 2) and are requested to proceed into the post-treatment phase.

# 7.1.2. Temporary Discontinuation from Study Treatment

Not applicable.

# 7.1.3. Discontinuation of Inadvertently Enrolled Patients

If the sponsor or investigator identifies a patient who did not meet enrollment criteria and was inadvertently enrolled, a discussion must occur between the sponsor CRP/CRS and the investigator to determine if the patient may continue in the study. If both agree it is medically appropriate to continue, the investigator must obtain documented approval from the sponsor

CRP/CRS to allow the inadvertently enrolled patient to continue in the study with or without treatment with investigational product.

# 7.1.4. Permanent Discontinuation from the Study

Some possible reasons that may lead to permanent discontinuation include:

- Enrollment in any other clinical trial involving an investigational product or enrollment in any other type of medical research judged not to be scientifically or medically compatible with this study
- Participation in the study needs to be stopped for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and good clinical practice (GCP)
- Investigator Decision
  - o the investigator decides that the patient should be discontinued from the study
  - o if the patient, for any reason, requires treatment with another therapeutic agent that has been demonstrated to be effective for the study indication (prevention of migraine) during Study Period III, discontinuation from the study occurs prior to introduction of the new agent
- Subject Decision
  - o the patient asks to be withdrawn from the study

Patients who discontinue the study early will have end-of-study (early termination) procedures performed as shown in the Schedule of Activities (Appendix 2) and are requested to proceed into the post-treatment phase.

# 7.1.5. Patients Lost to Follow-Up

A patient will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. Site personnel are expected to make diligent attempts to contact patients who fail to return for a scheduled visit or were otherwise unable to be followed up by the site.

# 8. Study Assessments and Procedures

Appendix 2 lists the Schedule of Activities, with the study procedures and their timing (including tolerance limits for timing).

Appendix 3 lists the laboratory tests that will be performed for this study.

Appendix 4 lists the tests that may be obtained in the event of a treatment-emergent hepatic abnormality.

Unless otherwise stated in the subsections below, all samples collected for specified laboratory tests will be destroyed within 60 days of receipt of confirmed test results. Certain samples may be retained for a longer period, if necessary, to comply with applicable laws, regulations, or laboratory certification standards.

# 8.1. Efficacy Assessments

# 8.1.1. Primary Efficacy Assessments

<u>ePRO Diary</u>: Patients will be asked to use an ePRO device (starting at Visit 2) to record headache symptoms, duration, and severity. The device also will be used to collect the name and dose of concomitant medications used for the acute treatment of migraine, and the use of other pain medications.

# 8.1.2. Secondary Efficacy Assessments

# 8.1.2.1. Patient Global Impression of Severity

The Patient Global Impression of Severity (PGI-S) scale (Guy 1976) is a patient-rated instrument that measures baseline illness severity. The PGI-S includes a range of possible responses, from 1 ("normal, not at all ill") to 7 ("extremely ill").

# 8.1.2.2. Patient Global Impression of Improvement

The Patient Global Impression of Improvement (PGI-I) scale (Guy 1976) is a patient-rated instrument that measures improvement of the patient's symptoms. It is a 7-point scale in which a score of 1 indicates the patient is "very much better," a score of 4 indicates the patient has experienced "no change," and a score of 7 indicates the patient is "very much worse."

# 8.1.3. Appropriateness of Assessments

All efficacy and safety assessments have been well documented and are generally regarded as reliable, accurate, and relevant in this patient population. This includes health outcomes measures considered to be appropriate for evaluating changes in quality of life, global functioning, and disability (Section 8.9).

#### 8.2. Adverse Events

Investigators are responsible for monitoring the safety of patients who have entered this study and for alerting Lilly or its designee to any event that seems unusual, even if this event may be considered an unanticipated benefit to the patient.

The investigator is responsible for the appropriate medical care of patients during the study.

Investigators must document their review of each laboratory safety report.

The investigator remains responsible for following, through an appropriate health care option, AEs that are serious or otherwise medically important, considered related to the investigational product or the study, or that caused the patient to discontinue the investigational product before completing the study. The patient should be followed until the event resolves, stabilizes with appropriate diagnostic evaluation, or is reasonably explained. The frequency of follow-up evaluations of the AE is left to the discretion of the investigator.

Lack of drug effect is not an AE in clinical studies, because the purpose of the clinical study is to establish treatment effect.

After the ICF is signed, study site personnel will record via eCRF the occurrence and nature of each patient's pre-existing condition(s), including clinically significant signs and symptoms of the disease under treatment in the study. In addition, site personnel will record via eCRF any change in the condition(s) and any new condition(s) as AEs. Investigators should record their assessment of the potential relatedness of each AE to protocol procedure or investigational product via eCRF.

The investigator will decide whether he or she interprets the observed AEs as reasonably possibly related to migraine headache, to the investigational product, study device, study procedure, or other concomitant treatment or pathologies.

The investigator will answer yes/no when making this assessment.

Planned surgeries and nonsurgical interventions should not be reported as AEs unless the underlying medical condition has worsened during the course of the study.

If a patient's investigational product is discontinued as a result of an AE, study site personnel must report this to Lilly or its designee via eCRF, clarifying if possible, the circumstances leading to discontinuations of treatment.

#### 8.2.1. Serious Adverse Events

An SAE is any AE from this study that results in one of the following outcomes:

- death
- initial or prolonged inpatient hospitalization
- a life-threatening experience (that is, immediate risk of dying)
- persistent or significant disability/incapacity

- congenital anomaly/birth defect
- considered significant by the investigator for any other reason: important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious, based upon appropriate medical judgment
- when a condition related to the investigational device (for example, prefilled syringe) necessitates medical or surgical intervention to preclude either permanent impairment of a body function or permanent damage to a body structure, the serious outcome of "required intervention" will be assigned

Although all AEs after signing the ICF are recorded in the eCRF, SAE reporting begins after the patient has signed the ICF and has received investigational product. However, if an SAE occurs after signing the ICF, but prior to receiving investigational product, it needs to be reported ONLY if it is considered reasonably possibly related to study procedure.

Study site personnel must alert Lilly or its designee of any SAE within 24 hours of investigator awareness of the event via a sponsor-approved method. If alerts are issued via telephone, they are to be immediately followed with official notification on study-specific SAE forms. This 24-hour notification requirement refers to the initial SAE information and all follow-up SAE information.

Pregnancy (during maternal or paternal exposure to investigational product) does not meet the definition of an AE. However, to fulfill regulatory requirements, any pregnancy that occurs during the study, including those in which conception occurred within 5 months after last administration of investigational product, should be reported using the SAE process to collect data on the outcome for both mother and fetus.

Investigators are not obligated to actively seek AEs or SAEs in patients once they have discontinued and/or completed the study (the patient summary eCRF has been completed). However, if the investigator learns of any SAE, including a death, at any time after a patient has been discharged from the study, and he/she considers the event reasonably possibly related to the study treatment or study participation, the investigator must promptly notify Lilly.

#### 8.2.1.1. Suspected Unexpected Serious Adverse Reactions

Suspected unexpected serious adverse reactions (SUSARs) are serious events that are not listed in the IB and that the investigator identifies as related to investigational product or procedure. United States 21 CFR 312.32 and European Union Clinical Trial Directive 2001/20/EC and the associated detailed guidance or national regulatory requirements in participating countries require the reporting of SUSARs. Lilly has procedures that will be followed for the recording and expedited reporting of SUSARs that are consistent with global regulations and the associated detailed guidance.

## 8.2.1.2. Adverse Event Monitoring with a Systematic Questionnaire

Suicidality will be assessed as required by the US Food and Drug Administration's Division of Neurology for use in clinical trials involving all drugs for neurological indications. Before administering the C-SSRS) [Posner et al. 2011]), study site personnel will question the patient
about any change in the pre-existing condition(s) and the occurrence and nature of any AEs. Nonserious AEs obtained through the questionnaire are recorded and analyzed separately. Only *serious* AEs and AEs leading to discontinuation elicited through the C-SSRS are to be recorded as AEs via eCRF. Serious adverse events must be reported to Lilly or its designee within 24 hours as SAEs. Any suicidal behavior, or suicidal ideation per items 4 or 5 (active suicidal ideation with some intent to act, either without specific plan or with specific plan and intent) would prompt referral of the patient to a mental health professional.

### 8.2.2. Complaint Handling

Lilly collects product complaints on investigational products and drug delivery systems used in clinical studies in order to ensure the safety of study participants, monitor quality, and to facilitate process and product improvements.

Patients will be instructed to contact the investigator as soon as possible if he or she has a complaint or problem with the investigational product (or drug delivery system such as a prefilled syringe) so that the situation can be assessed.

### 8.3. Treatment of Overdose

No data are available at this stage of development.

### 8.4. Safety Assessments

### 8.4.1. Electrocardiograms

For each patient, a single, 12-lead digital ECG will be collected at the visits shown in the Schedule of Activities (Appendix 2). Electrocardiograms will have a central overread and should be recorded according to the study-specific recommendations included in the ECG manual.

Any clinically significant findings from ECGs that result in a diagnosis should be reported to Lilly or its designee as an AE via eCRF.

# 8.4.2. Vital Signs

Vital signs will include body temperature, blood pressure, and pulse. Blood pressure and pulse will be measured in triplicate in the sitting position prior to blood draws and study drug administration (see Study Schedule [Appendix 2]).

Any clinically significant findings from vital signs measurement that result in a diagnosis should be reported to Lilly or its designee as an AE via eCRF.

# 8.4.3. Laboratory Tests

For each patient, laboratory tests detailed in Appendix 3 should be conducted according to the Schedule of Activities (Appendix 2).

Any clinically significant findings from laboratory tests that result in a diagnosis should be reported to Lilly or its designee as an AE via eCRF.

In addition, an immunogenicity plasma sample will be collected, when possible, for any patient who experiences a potential systemic allergic/hypersensitivity reaction during the study as judged by the investigator. This immunogenicity plasma sample should be collected immediately or as soon as possible, taking into consideration the availability and wellbeing of the patient. Exact date and time of the sample should be recorded on the laboratory requisition form.

#### 8.4.4. Other Tests

Not applicable.

### 8.4.5. Safety Monitoring

Investigators are responsible for monitoring individual patient safety throughout the trial. If a study patient/subject experiences elevated ALT  $\geq$ 3X ULN, ALP  $\geq$ 2X ULN, or elevated TBL  $\geq$ 2X ULN, clinical and laboratory monitoring should be initiated by the investigator. Details for hepatic monitoring depend upon the severity and persistence of observed laboratory test abnormalities. To ensure patient/subject safety and comply with regulatory guidance, the investigator is to consult with the Lilly CRP/CRS regarding collection of specific recommended clinical information and follow-up laboratory tests. See Appendix 4.

Neurological examinations will be conducted at screening, Month 3 and Month 6 of treatment, as well as at the final visit of the follow-up period or early termination visit in order to assess for any signs of pre-existing or treatment-emergent neurological abnormalities such as stroke or other cerebrovascular events. If a study patient experiences signs of a cerebrovascular event, appropriate follow-up and clinical management should be conducted by the investigator, and the Lilly CRP/CRS should be consulted regarding collection of further clinical information and follow-up testing.

Lilly will periodically review evolving aggregate safety data within the study by appropriate blinded methods. In addition, safety data for the trial will also be reviewed periodically by an independent Data Monitoring Committee (DMC; an advisory group for this study formed to protect the integrity of data; refer to Interim Analyses section [Section 9.8]). In the event that safety monitoring uncovers an issue that needs to be addressed by unblinding at the group level, members of the DMC can request additional analyses of the safety data.

### 8.5. Pharmacokinetics

At the visits and times specified in the Schedule of Activities (Appendix 2), venous blood samples of approximately 2.5 mL each will be collected to determine the serum concentrations of LY2951742. A maximum of 3 samples may be collected at additional time points during the study if warranted and agreed upon between both the investigator and sponsor. Instructions for the collection and handling of blood samples will be provided by the sponsor.

When a blood sample is collected, the time and date of last dose administration prior to blood sampling should be recorded. The actual date and time (24-hour clock time) of each sampling will be recorded. LY2951742 concentration information that may/would unblind the study will

not be reported to investigative sites or blinded personnel until the study has been unblinded. Bioanalytical samples collected to measure investigational product concentration will be retained for a maximum of 1 year following last patient visit for the study.

A validated assay will be used to determine serum LY2951742 concentrations. Samples will be analyzed at a laboratory approved by the sponsor.

It is intended that blood samples collected from patients who received placebo should not be analyzed for determination of serum concentrations of LY2951742.

### 8.6. Pharmacodynamics

At the visits and times specified in the Schedule of Activities (Appendix 2), venous blood samples will be collected to determine the plasma concentrations of CGRP. A maximum of 3 samples may be collected at additional time points during the study if warranted and agreed upon between both the investigator and sponsor. Instructions for the collection and handling of blood samples will be provided by the sponsor. When a blood sample is collected, the time and date of last dose administration prior to blood sampling should be recorded. The actual date and time (24-hour clock time) of each sampling will be recorded.

A validated LY2951742-tolerant assay will be used to determine plasma CGRP concentrations. Samples will be analyzed at a laboratory approved by the sponsor.

Plasma CGRP concentration information that may/would unblind the study will not be reported to investigative sites or blinded personnel until the study has been unblinded.

Bioanalytical samples collected to measure CGRP will be identified by the patient number (coded) and retained for a maximum of 1 year following last patient visit for the study at a facility selected by the sponsor.





### 8.8. Biomarkers

Blood samples for non-genetic biomarker research will be collected at the times specified in the Schedule of Activities (Appendix 2), where local regulations and ERBs allow.

Samples will be used for research on the drug target, disease process, pathways associated with migraine headache and/or other pain conditions, mechanism of action of LY2951742, and/or research method or in validating diagnostic tools or assay(s) related to migraine headache and/or other pain conditions.

All biomarker samples will be coded with the patient number. These samples and any data generated can be linked back to the patient only by the investigator site personnel. Samples will be destroyed according to a process consistent with local regulations.

Samples will be retained for a maximum 15 years after the last patient visit for the study, or for a shorter period if local regulations and ERBs impose shorter time limits, at a facility selected by the sponsor. This retention period enables use of new technologies, response to regulatory questions, and investigation of variable response that may not be observed until later in drug development or when the drug is commercially available.

# 8.8.1. Samples for Immunogenicity Research

Where local regulations and ERBs allow, blood samples for immunogenicity testing will be collected to determine antibody production against LY2951742 as specified in the Schedule of Activities (Appendix 2). Immunogenicity will be assessed by a validated assay designed to detect anti-drug antibodies in the presence of the investigational product. Antibodies may be further characterized and/or evaluated for their ability to neutralize the activity of LY2951742.

Samples will be retained for a maximum of 15 years after the last patient visit for the study, or for a shorter period if regulations and ERBs impose shorter time limits, at a facility selected by the sponsor. The duration allows the sponsor to respond to future regulatory requests related to LY2951742.

### 8.9. Health Economics

Health economic, disability and quality of life assessments of LY2951742 in patients with migraine will be based on the following scales:

Migraine Disability Assessment test (MIDAS): The MIDAS was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that

reflect the number of days reported as missing, or with reduced productivity at work or home and social events; a higher value is indicative of more disability (Stewart 1999; Stewart 2001). This instrument is considered highly reliable and valid; and is correlated with clinical judgment regarding the need for medical care (Stewart 1999; Stewart 2001).

Migraine Specific Quality of Life questionnaire (MSQ v2.1): The MSQ v2.1 is a self-administered health status instrument, and was developed to address physical and emotional limitations of specific concern to individuals suffering from migraine headaches. The instrument consists of 14 items that address 3 domains: (1) Role Function-Restrictive; (2) Role Function-Preventive; and, (3) Emotional Function (Jhingran 1998). The instrument was designed with a 4-week recall period, and is considered reliable, valid and sensitive to change in migraine (Jhingran 1998; Rendas-Baum 2013). Clinically meaningful differences for each domain have been established and are widely used in the literature.

# 9. Statistical Considerations and Data Analysis

### 9.1. Determination of Sample Size

The study will enroll approximately 825 patients. Eligible patients will be randomized in blinded fashion in a 2:1:1 ratio to placebo (target of 413 patients), LY2951742 120 mg/month (target of 206 patients), or 240 mg/month (target of 206 patients). With the assumption of a 26% discontinuation rate and an effect size of 0.33, it is estimated that this sample size will provide approximately 95% power that at least 1 dose of LY2951742 will separate from placebo at a two-sided significance level of 0.05 based on simulations using Dunnett (Dunnett 1955) test. Assumptions in the simulations were based on data from two double-blind, placebo-controlled, Phase 2 studies, with adjustment to reflect the longer treatment duration and greater variability expected in a larger, multi-country Phase 3 study.

Approximately 100 sites in 11 countries are planned for inclusion in Study CGAH, with an average of approximately 8 patients to be randomized at each investigative site. The final number of sites, countries, and patients per site may vary depending on sites' enrollment rates. Approximately 1557 patients may be screened to ensure randomization of 825 patients, with an estimated 611 patients completing the study.

### 9.2. General Statistical Considerations

Statistical analysis of this study will be the responsibility of Lilly or its designee. Details of statistical analysis methods will be described in the statistical analysis plan (SAP) document.

Unless otherwise specified, analyses will be conducted on an intent-to-treat (ITT) population, which will include all patients who are randomized and receive at least one dose of investigational product. Patients in the ITT population will be analyzed according to the treatment group to which they are randomized. When change from baseline is assessed, the patient will be included in the analysis only if he/she has a baseline and a postbaseline measurement.

The primary analysis will be performed using a restricted maximum likelihood-based mixed models repeated measures (MMRM) technique with prespecified model terms (Section 9.4.1).

Visitwise binary efficacy variables will be analyzed using a generalized linear mixed model (GLIMMIX) as pseudo-likelihood-based mixed effects repeated measures analysis.

In addition to the MMRM approach, analysis of covariance (ANCOVA) model or analysis of variance (ANOVA) with the last observation carried forward (LOCF) will also be implemented. When an ANCOVA model is used to analyze a continuous variable, the model will contain the main effects of treatment and region, as well as the continuous fixed covariates of baseline. The ANOVA model will use the same terms except the continuous fixed covariate of baseline. Type III sum-of-squares for the least-squares means will be used for the statistical comparisons.

Continuous efficacy and health outcome endpoints will be analyzed using MMRM methods, as well as an ANCOVA model with LOCF imputation if deemed appropriate.

Categorical comparisons between treatment groups will be performed using Cochran-Mantel-Haenszel (CMH) controlling for region or using the Fisher's exact test, where appropriate.

Patients will be pooled within each region for statistical analysis purposes. Region will be defined in the SAP.

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, unless otherwise stated.

Any change to the data analysis methods described in the protocol will require an amendment ONLY if it changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol, and the justification for making the change, will be described in the clinical study report or SAP. Changes may only be made in the SAP prior to unblinding. Additional exploratory analyses of the data will be conducted as deemed appropriate.

### 9.3. Treatment Group Comparability

# 9.3.1. Patient Disposition

The number and percentage of ITT patients who complete the study or discontinue early will be summarized for all treatment groups for Study Period III (double-blind treatment) and Study Period IV (post-treatment follow-up) both overall and by visit.

Patient allocation by investigator will be summarized for Study Period III for all ITT patients. Patient allocation by investigator will also be listed for all study periods.

#### 9.3.2. Patient Characteristics

The following patient characteristics at baseline will be summarized by treatment group for all ITT patients:

- Demographic (age, gender, ethnic origin, height, weight, body mass index)
- Migraine headache, headache, variation of migraine/headache measures per 30-day baseline period.
- Alcohol, tobacco, caffeine and nicotine consumption
- Medical history and pre-existing condition

Medical history and pre-existing conditions will be summarized by preferred term within system organ class (SOC).

# 9.3.3. Concomitant Therapy

The proportion of patients who received concomitant medication (as recorded via eCRF) as well as abortive medications (recorded through ePRO) will be summarized for all ITT patients for Study Period III and Study Period IV separately.

# 9.3.4. Treatment Compliance

Not applicable.

### 9.3.5. Electronic Patient-reported Outcome Diary Compliance

ePRO diary compliance at each period (including baseline, Month 1, 2, 3, ... till Month 10) will be calculated. Diary compliance at each period is calculated as:

Actual number of diary days in the period Expected number of diary days in the period \* 100

Actual number of diary days is calculated as the total number of days with non-missing answers.

### 9.4. Primary and Secondary Analyses

### 9.4.1. Primary Analyses

The primary efficacy measure is the overall mean change from the baseline period in the number of monthly migraine headache day during the 6-month double-blind treatment phase, and the primary analysis will evaluate the efficacy of LY2951742 (120 or 240 mg/month) compared with placebo.

The primary analysis will be performed using a restricted maximum likelihood-based MMRM technique. The analysis will include the fixed categorical effects of treatment, region, month, and treatment-by-month interaction, as well as the continuous fixed covariates of baseline number of migraine headache days and baseline number of migraine headache days-by-month interaction.

An unstructured covariance structure will be used to model within-patient errors. The Kenward-Roger (Kenward and Roger 1997) approximation will be used to estimate denominator degrees of freedom. If the model does not converge with both the Hessian and the G matrix being positive definite under the default fitting algorithm used by PROC MIXED, the Fisher scoring algorithm will be implemented by specifying the SCORING option in SAS. If the model still fails to converge, the model will be fit using covariance matrices of the following order specified by a decreasing number of covariance parameters until convergence is met:

- Heterogeneous Toeplitz
- Heterogeneous First-order autoregressive
- Toeplitz
- First-order autoregressive

When the unstructured covariance matrix is not utilized, the sandwich estimator (Diggle and Kenward 1994) will be used to estimate the standard errors of the fixed effects parameters. The sandwich estimator is implemented by specifying the EMPIRICAL option in SAS<sup>®</sup>. When the sandwich estimator is utilized, the Kenward-Roger approximation for denominator degrees of freedom cannot be used. Instead, the denominator degrees of freedom will be partitioned into between-subject and within-subject portions by the DDFM=BETWITHIN option in SAS<sup>®</sup>. SAS<sup>®</sup> PROC MIXED will be used to perform the analysis.

# 9.4.2. Key Secondary Analyses

The key secondary objectives (see Table CGAH.1) will be tested using an appropriate multiple testing approach providing strong control of the familywise error rate (for the primary and key secondary tests) at a one-sided 0.025 alpha level (or, equivalently, two-sided 0.05 alpha level).





There will be no adjustments for multiplicity for analyses of other endpoints. If the multiple testing approach for key secondary measures only needs to be changed, the updated approach will be provided in the SAP, and it should not lead to modification of this protocol.

The key secondary measures will be analyzed for the double-blind treatment (Study Period III).

For the continuous key secondary measures, the change from baseline during the 6-month double-blind treatment phase will be analyzed from repeated measures analyses as described in Section 9.4.1. For the analysis of 50%, 75%, and 100% response, the percentage of patients meeting response criteria during the 6-month double-blind treatment phase will be estimated for each treatment from a categorical, pseudo-likelihood-based repeated measures analysis of longitudinal binary outcomes indicating whether patients meet response criteria.

This analysis will be implemented using the GLIMMIX procedure in SAS.

# 9.4.3. Other Secondary and Tertiary Efficacy Analyses

The other secondary and exploratory efficacy analyses will be conducted for the double-blind treatment phase, and for the double-blind treatment and post-treatment follow-up phases (Study Period III and Study Period IV) combined. Further details regarding other secondary and tertiary efficacy analyses are summarized in the SAP.

### 9.5. Safety Analyses

The safety analyses will be conducted for the double-blind treatment and post-treatment follow-up phases, as well as the two periods combined. For the two phases combined, only repeated measures and time-to-event analyses will be conducted.

The safety and tolerability of treatment will be assessed by summarizing the following:

- adverse events
  - o treatment-emergent adverse events (TEAEs)
    - by preferred term
    - by SOC
    - by maximum severity
    - by outcome
    - considered to be related to investigational product by investigator
  - serious adverse event
  - o adverse event leading to discontinuation
- Suicidal ideation and behaviors assessed by solicited questioning using the C-SSRS
- Vital signs and weight
- electrocardiograms
- Laboratory measurements
- Anti-LY2951742 antibody

# 9.5.1. Categorical Safety Variables

Unless specified otherwise, the categorical safety analyses will include both schedule and unscheduled visits.

Comparisons between treatment groups for all categorical safety measures will be made using the Fisher's exact test for Study Period III (double-blind treatment) with the ITT population. Descriptive statistics only will be presented for the treatment groups in the post-treatment follow-up phase (Study Period IV) with the post-treatment population.

#### 9.5.2. Adverse Events

Treatment-emergent adverse events are defined as the reported AEs that first occurred or worsened during the postbaseline phase compared with baseline phase. For each TEAE, the severity level of the event (mild, moderate, or severe) will be determined by patient or physician opinion. The Medical Dictionary for Regulatory Activities (MedDRA) Lowest Level Term will be used in the treatment-emergent computation. For each Lowest Level Term, the maximum severity at baseline will be used as the baseline severity. If the maximum severity during

postbaseline is greater than the maximum baseline severity, the event is considered to be treatment-emergent for the specific postbaseline period. For each patient and TEAE, the maximum severity for the MedDRA level being displayed (PT, High Level Term, or SOC) is the maximum postbaseline severity observed from all associated Lowest Level Terms mapping to that MedDRA level.

For events that are gender-specific, the denominator and computation of the percentage will include only patients from the given gender.

### 9.5.3. Suicide-Related Thoughts and Behaviors

Suicidal ideation, suicidal behavior, and non-suicidal self-injurious behavior based on the C-SSRS will be summarized by treatment group. For each of the following events, the number and percentage of patients with the event will be enumerated by treatment: completed suicide, non-fatal suicide attempt, interrupted attempt, aborted attempt, preparatory acts or behavior, active suicidal ideation with specific plan and intent, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with any methods (not plan) without intent to act, non-specific active suicidal thoughts, wish to be dead, and non-suicidal self-injurious behavior. In addition, the number and percentage of patients who experienced at least one of the composite measures during Study Period III and Study Period IV separately will be presented and compared. These include suicidal acts (completed suicide and nonfatal suicidal attempts), suicidal behavior (suicidal acts, interrupted attempts, aborted attempts, and preparatory acts or behavior), treatment-emergent suicidal ideation or treatment-emergent suicidal behavior.

The Fisher's exact test will be used for treatment comparisons.

# 9.5.4. Vital Signs and Weight

Vital signs collected during the study include systolic and diastolic blood pressure, pulse, and temperature. Blood pressure and pulse measurements will be taken when the patient is in a sitting position. Three measurements of sitting blood pressure and pulse will be collected at every visit; the 3 sitting blood pressure and pulse measurements will be averaged and used as the value for that visit for analysis.

The incidence rates of patients with treatment-emergent vital sign and weight changes based at any time postbaseline and at LOCF endpoint will be assessed using the Fisher's exact test. Specific criteria for treatment emergent definition will be documented in the SAP.

# 9.5.5. Electrocardiogram Intervals and Heart Rate

Analyses of corrected QT interval will be calculated using two correction formulas. The QTcF (measured in milliseconds [msec]) will be calculated with Fridericia's formula as QT/RR <sup>1/3</sup>. The Large Clinical Trial Population Based QT Correction (QTcLCTPB) (msec) will be calculated with the formula as QT/RR <sup>0.413</sup>. The number and percent of patients meeting criteria for treatment-emergent abnormalities in ECG intervals (pulse rate [PR], QRS, QTcF, and QTcLCTPB) and heart rate at any time during study will be summarized. Treatment group comparisons will be performed using the Fisher's exact test.

### 9.5.6. Laboratory Tests

The incidence rates of patients with treatment-emergent abnormal, high, or low laboratory values at any time postbaseline and at LOCF endpoint will be assessed using the Fisher's exact test for each laboratory test.

Patients will be defined as having a treatment-emergent low value if they have all normal or high values at baseline, followed by a value below the lower reference limit at any postbaseline visit. Patients with all normal or high values at baseline (no low values) will be included in the analysis of treatment-emergent low laboratory values. Patients will be defined as having a treatment-emergent high value if they have all normal or low values at baseline, followed by a value above the upper reference limit at any postbaseline visit. Patients with all normal or low values at baseline (no high values) will be included in the analysis of treatment-emergent high laboratory values.

For analytes simply classified as normal or abnormal, patients will be defined as having a treatment-emergent abnormal value if they have all normal values at baseline, followed by an abnormal value at any postbaseline visit. Patients with all normal values at baseline will be included in the analysis of treatment-emergent abnormal laboratory values.



# 9.7. Other Analyses

### 9.7.1. Health Economics

The change from baseline to each postbaseline visit for the double-blind treatment phase and for the double-blind treatment and post-treatment follow-up phases combined for MSQ v2.1 (Role Function-Restrictive, Role Function-Preventive, Emotional Function, and total score) and MIDAS (item scores and total score) will be analyzed. In addition, categorical analysis for the frequency measure will be performed.

# 9.7.2. Subgroup Analyses

Subgroup analyses will be performed for the primary efficacy measure (change from baseline in the number of migraine headache days) separately for each of the subgroup populations listed in Table CGAH.4. Subgroup analyses will be conducted only for the ITT patients in Study Period III

Each of the subgroup analyses for the primary measure of change from baseline in the number of migraine headache days will be conducted using MMRM. The same MMRM model described in Section 9.4.1 will be used, with terms of subgroup, subgroup-by-treatment, subgroup-by-month, and subgroup-by-treatment-by-month interactions added as additional co variates.

Table CGAH.4. Definition of Subgroup Variables

| Subgroup Variable | Categories |
|---|---|
| • Sex | Male, female |
| Racial Origin (combine those with | American Indian / Alaskan Native |
| less than 10%) | Asian |
| | Black / African American |
| | Native Hawaiian / Pacific Islander |
| | White |
| | Multiple |
| • Ethnicity | Hispanic or Latino |
| | Not Hispanic or Latino |
| Region | Defined in the statistical analysis plan (SAP) |
| Baseline number of migraine | 2 levels of baseline migraine frequency : |
| headache days | • <8 migraine headache days |
| | • ≥8 migraine headache days |
| Treatment-resistant status | Treatment-resistant status about whether a patient has failed 2 or |
| | more prophylactic treatments (Yes or No) |
| Having aura or not (during baseline) | Yes or No |
| period) | |
| Baseline anti-drug antibody status | Any confirmed positive anti-drug antibody at baseline (Yes |
| | versus No) |
| Neutralizing anti-drug antibody | Any positive neutralizing anti-drug antibody time point (Yes |
| status | versus No) – note that neutralizing ADA assays are performed |
| | only on confirmed-positive anti-drug antibodies. |
| Treatment-emergent anti-drug | Any treatment-emergent anti-drug antibody (Yes versus No) |
| antibody status | |

# 9.8. Interim Analyses

Two interim analyses are anticipated for this study. The first possible interim analysis will occur during Study Period III (double-blind treatment) and could result in stopping the trial for safety or futility. This analysis is planned to occur when approximately 330 (40% of the total sample size) randomized patients have had the chance to complete at least 3 months of the treatment period. The interim analysis will be conducted by an independent data monitoring committee (DMC) with members external to Lilly. The data from the interim analysis will be used to evaluate whether to stop or modify the study for futility and/or safety issues. Stopping rules for futility at this interim analysis will be based on the conditional power of comparing LY2951742 to placebo. Specifically, conditional power represents the probability that the ongoing trial will

result in a statistically significant difference between LY2951742 and placebo at end of the trial, based on the data available at the time of the interim analysis. Rules for stopping the study are detailed in the Statistical Analysis Center SAP and the DMC Charter. Only the DMC is authorized to evaluate unblinded interim efficacy and safety analyses. Study sites will receive information about interim results ONLY if they need to know for the safety of their patients. There is no inflation of type 1 error due to the conduct of a futility analysis (Snapinn et al. 2006), so no adjustment to the nominal significance level will be made for the primary analysis as a result of a futility assessment.

The second interim analysis will be conducted after all patients have had the opportunity to complete Study Period III, and thus, will be the final analysis of the primary efficacy endpoint.

Unblinding details are specified in the unblinding plan section of the SAP or a separate unblinding plan document.

Additional interim analyses may be conducted in support of regulatory submissions if necessary.

# 10. Study Governance Considerations

# 10.1. Regulatory and Ethical Considerations, Including the Informed Consent Process

### 10.1.1. Informed Consent

The investigator is responsible for ensuring:

- that the patient understands the potential risks and benefits of participating in the study
- that informed consent is given by each patient. This includes obtaining the appropriate signatures and dates on the ICF prior to the performance of any protocol procedures and prior to the administration of investigational product.
- answering any questions the patient may have throughout the study and sharing in a timely manner any new information that may be relevant to the patient's willingness to continue his or her participation in the trial.

### 10.1.2. Ethical Review

The investigator must give assurance that the ERB was properly constituted and convened as required by International Conference on Harmonisation (ICH) guidelines and other applicable laws and regulations.

Documentation of ERB approval of the protocol and the ICF must be provided to Lilly before the study may begin at the investigative site(s). Lilly or its representatives must approve the ICF, including any changes made by the ERBs, before it is used at the investigative site(s). All ICFs must be compliant with the ICH guideline on GCP.

The study site's ERB(s) should be provided with the following:

- the current IB and updates during the course of the study
- informed consent document
- relevant curricula vitae

# 10.1.3. Regulatory Considerations

This study will be conducted in accordance with:

- consensus ethics principles derived from international ethics guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
- applicable ICH GCP guidelines
- applicable laws and regulations

Some of the obligations of the sponsor will be assigned to a third-party organization (TPO).

### 10.1.4. Investigator Information

Investigators in this clinical trial should be neurologists, headache specialists, or other specialists with experience in headache clinical trials and treating migraine headache patients.

### 10.1.5. Protocol Signatures

The sponsor's responsible medical officer will approve the protocol, confirming that, to the best of his or her knowledge, the protocol accurately describes the planned design and conduct of the study.

After reading the protocol, each principal investigator will sign the protocol signature page and send a copy of the signed page to a Lilly representative.

# 10.1.6. Final Report Signature

The clinical study report (CSR) coordinating investigator will sign the final CSR for this study, indicating agreement that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

An investigator selected by the study team will serve as the CSR coordinating investigator. If this investigator is unable to fulfill this function, another investigator will be chosen by Lilly to serve as the CSR coordinating investigator.

The sponsor's responsible medical officer and statistician will approve the final CSR for this study, confirming that, to the best of his or her knowledge, the report accurately describes the conduct and results of the study.

# 10.2. Data Quality Assurance

To ensure accurate, complete, and reliable data, Lilly or its representatives will do the following:

- provide instructional material to the study sites, as appropriate
- sponsor start-up training to instruct the investigators and study coordinators. This
  training will give instruction on the protocol, the completion of the eCRFs, and
  study procedures.
- make periodic visits to the study site
- be available for consultation and stay in contact with the study site personnel by mail/e-mail, telephone, and/or fax
- review and evaluate eCRF data and use standard computer edits to detect errors in data collection
- conduct a quality review of the database

In addition, Lilly or its representatives will periodically check a sample of the patient data recorded against source documents at the study site. The study may be audited by Lilly or its representatives, and/or by regulatory agencies at any time. Investigators will be given notice before an audit occurs.

To ensure the safety of participants in the study, and to ensure accurate, complete, and reliable data, the investigator will keep records of ECGs, laboratory tests, clinical notes, and patient medical records in the patient files as original source documents for the study according to retention requirements as outlined by the ICH guidelines. If requested, the investigator will provide the sponsor, applicable regulatory agencies, and applicable ERBs with direct access to original source documents.

### 10.2.1. Data Capture System

An electronic data capture system will be used in this study. The site maintains a separate source for the data entered by the site into the sponsor-provided electronic data capture system.

Some or all of a patient's data will be directly entered into the eCRF at the time the information is obtained. In instances where direct data entry is not used, the site will maintain source documentation in the trial files, and the patient's data will be transcribed into the eCRF. Any data for which the eCRF will serve as the source document, or any other data not entered directly into the eCRF, will be identified and documented by the site in the site's trial file. For data handled by a data management TPO, eCRF data and some or all data that are related will be managed and stored electronically in the TPO system. Subsequent to the final database lock, validated data will be transferred to the sponsor. For data handled internally, eCRF data and some or all data that are related will be managed by the sponsor and stored electronically in the sponsor's system.

In this study, patient migraine headache data will be collected directly via an ePRO diary as part of an ePRO/Clinical Outcome Assessment (COA) system. Patient-rated scales/questionnaires will be collected directly via an ePRO tablet device at each visit. Data entered into the ePRO/COA system will serve as the source data.

If ePRO/COA records are stored at a third-party site, investigator sites will have continuous access to the source documents during the study and will receive an archival copy at the end of the study for retention.

Any data for which the ePRO/COA instrument record will serve to collect source data will be identified and documented by each site in that site's study file.

Case report form data will be encoded and stored in a clinical trial database. Data managed by a central vendor, such as laboratory test data or ECG data, will be stored electronically in the central vendor's database system. Data will subsequently be transferred from the central vendor to the Lilly data warehouse. Data from complaint forms submitted to Lilly will be encoded and stored in the global product complaint management system.

# 10.3. Study and Site Closure

# 10.3.1. Discontinuation of Study Sites

Study site participation may be discontinued if Lilly or its designee, the investigator, or the ERB of the study site judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

# 10.3.2. Discontinuation of the Study

The study will be discontinued if Lilly or its designee judges it necessary for medical, safety, regulatory, or other reasons consistent with applicable laws, regulations, and GCP.

### 11. References



Diggle P, Kenward MG. Informative drop-out in longitudinal data analysis. *J Royal Statist Soc Series C: Appl Statist*. 1994;43(1):49-93.



- Goadsby PJ, Edvinsson L. The trigeminovascular system and migraine: Studies characterizing cerebrovascular and neuropeptide changes seen in humans and cats. *Ann Neurol*. 1993;33(1):48-56.
- Goadsby PJ, Edvinsson L, Ekman R. Vasoactive peptide release in the extracerebral circulation of humans during migraine headache. *Ann Neurol*. 1990;28(2):183-187.
- Guy W. ECDEU assessment manual for psychopharmacology, revised 1976. Rockville, MD: National Institute of Mental Health, Psychopharmacology Research Branch. p 217-222. Available at: https://archive.org/details/ecdeuassessmentm1933guyw. Accessed January 11, 2016.



- [ICHD-3] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). *Cephalalgia*. 2013;33(9):629-808.
- Jhingran P, Osterhaus JT, Miller DW, Lee JT, Kirchdoetfer L. Development and validation of the migraine-specific quality-of-life questionnaire. *Headache*. 1998;38(4):295-302.
- Kenward MG, Roger JH. Small sample inference for fixed effects from restricted maximum likelihood. *Biometrics*. 1997;53(3):983-997.

# CCI

- Lassen LH, Haderslev PA, Jacobsen VB, Iversen HK, Sperling B, Olesen J. CGRP may play a causative role in migraine. *Cephalalgia*. 2002;22(1):54-61.
- Lassen LH, Jacobsen VB, Pedersen PA, Sperling B, Iversen H, Olesen J. Human calcitonin generelated peptide (hCGRP)-induced headache in migraineurs. *Eur J Neurol*. 1998;5(suppl 3):S63.

# CCI

Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial

- validity and internal consistency findings from three multisite studies with adolescents and adults. *Am J Psychiatry*. 2011;168(12):1266-1277.
- Rendas-Baum R, Bloudek LM, Maglinte GA, Varon SF. The psychometric properties of the Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ) in chronic migraine patients. *Qual Life Res.* 2013;22(5):1123–1133.
- Rizzoli P. Preventive pharmacotherapy in migraine. *Headache*. 2014;54(2):364-369.
- Silberstein SD, Holland S, Freitag F, Dodick DW, Argoff C, Ashman E. Evidence-based guideline update: Pharmacologic treatment for episodic migraine prevention in adults: Report of the Quality Standards Subcommittee of the American Academy of Neurology and the American Headache Society. Neurology. 2012;78(17):1337-1345.
- Snapinn S, Chen MG, Jiang Q, Koutsoukos T. Assessment of futility in clinical trials. *Pharm Stat.* 2006;5(4):273–281.
- Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability (abstract). Neurology . 2001;56 (6 Suppl 1):S20–S28.
- Stewart WF, Lipton RB, Kolodner K, Liberman J, Sawyer J. Reliability of the migraine disability assessment score in a population-based sample of headache sufferers. *Cephalalgia* 1999;19(2):107-114.
- Villalón CM, Olesen J. The role of CGRP in the pathophysiology of migraine and efficacy of CGRP receptor antagonists as acute antimigraine drugs. *Pharmacol Ther*. 2009;124(3):309-323.
- Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, et al. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. *Lancet*. 2012;380(9859): 2163-2196.

# Appendix 1. Abbreviations and Definitions

| Term | Definition |
|---|---|
| AE | adverse event: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. |
| complaint | A complaint is any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, purity, durability, reliability, safety or effectiveness, or performance of a drug or drug delivery system. |
| CRP/CRS | Lilly Clinical Research Physician/Clinical Research Scientist |
| enroll | The act of assigning a patient to a treatment. Patients who are enrolled in the trial are those who have been assigned to a treatment. |
| enter | Patients entered into a trial are those who sign the informed consent form directly or through their legally acceptable representatives. |
| ePRO | electronic patient-reported outcomes |
| interim analysis | An interim analysis is an analysis of clinical study data, separated into treatment groups, that is conducted before the final reporting database is created/locked. |
| investigational<br>product | A pharmaceutical form of an active ingredient or placebo being tested or used as a reference in a clinical trial, including products already on the market when used or assembled (formulated or packaged) in a way different from the authorized form, or marketed products used for an unauthorized indication, or marketed products used to gain further information about the authorized form. |
| ITT | intent to treat: The principle that asserts that the effect of a treatment policy can be best assessed by evaluating on the basis of the intention to treat a patient (that is, the planned treatment regimen) rather than the actual treatment given. It has the consequence that patients allocated to a treatment group should be followed up, assessed, and analyzed as members of that group irrespective of their compliance to the planned course of treatment. |
| IWRS | interactive web-response system |
| SAE | serious adverse event |
| TEAE | treatment-emergent adverse event: Any untoward medical occurrence that either occurs or worsens at any time after treatment baseline and that does not necessarily have to have a causal relationship with this treatment. |

# Appendix 2. Schedule of Activities

Schedule of Activities, Protocol I5Q-MC-CGAH

| Study Period (SP) | SP I-<br>Screening | SP II-<br>Prospective<br>Baseline | | SP III - Treatment | | | | | | | | | | | -up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (Target) Interval (days) since previous visit | | | 30-45 | 14 | 16 | 30 | 30 | 30 | 15 | 15 | 15 | 15 | 60 | 60 | |
| Allowable range (days)<br>between visits | 3-45 | 30-40 <sup>a</sup> | | | | | | | | | | | | | |
| Interval allowance (days) | | | | +/- 1 | +/- 3 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 5 | +/- 5 | ET |
| Visit | 1 | 2 | 3 | 4 <sup>b</sup> | 5 | 6 | 7 | 8 | 9° | 10 | 11° | 12 | 13 | 14 | |
| Month | | | 0 | 0.5 | 1 | 2 | 3 | 4 | 4.5 | 5 | 5.5 | 6 | 8 | 10 | |
| Assessments and Procedur | es | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | |
| Inclusion/exclusion | X | X | X | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Physical examination | X | | | | | | | | | | | | | | |
| Neurological examination <sup>d</sup> | X | | | | | | X | | | | | X | | X | X |
| Height | X | | | | | | | | | | | | | | |
| Weight | X | | | | | | | | | | | X | | X | X |
| Waist and hip circumference | X | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | |
| Pre-specified migraine history | | X | | | | | | | | | | | | | |

| Visit | 1 | 2 | 3 | 4 <sup>b</sup> | 5 | 6 | 7 | 8 | 9° | 10 | 11 <sup>c</sup> | 12 | 13 | 14 | ET |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month | | | 0 | 0.5 | 1 | 2 | 3 | 4 | 4.5 | 5 | 5.5 | 6 | 8 | 10 | |
| Substance use | X | | | | | | | | | | | | | | |
| ECGe | X | | X | | | | | | | | | X | | X | X |
| Vital signsf | X | | X | | X | X | X | X | | X | | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | | X | | X | X | X | X |
| Concomitant medications | X | X | X | | X | X | X | X | | X | | X | X | X | X |
| ePRO training | | X | | | | | | | | | | | | | |
| ePRO daily patient entries | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Patient training video | | | X | | | | | | | | | | | | |
| Clinical Laboratory Tests a | and Sampling | g Schedules | | | | | | | | | | | | | - |
| Hematology | X | | X | | | | X | | | | | X | | X | X |
| Clinical chemistry | X | | Xg | | | | Xg | | | | | Xg | | Xg | Xg |
| HDL | X | | Xg | | | | Xg | | | | | Xg | | Xg | Xg |
| HbA1c | | | X | | | | | | | | | X | | X | X |
| Fasting insulin/<br>fasting C-peptide | | | X <sup>g</sup> | | | | | | | | | $X^{g}$ | | | X <sup>g</sup> |
| Urinalysis <sup>h</sup> | X | | X | | | | | | | | | X | | X | X |
| Serum Pregnancy (for<br>women of childbearing<br>potential) or FSH at Visit<br>1 (all other female<br>patients) <sup>i</sup> | X | | | | | | | | | | | X | | X | X |
| Urine pregnancyi | | | X | | X | X | X | X | | X | | | | | |
| Urine drug screen | X | | | | | | | | | | | | | | |

| Visit | 1 | 2 | 3 | <b>4</b> <sup>b</sup> | 5 | 6 | 7 | 8 | 9° | 10 | 11° | 12 | 13 | 14 | ET |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month | | | 0 | 0.5 | 1 | 2 | 3 | 4 | 4.5 | 5 | 5.5 | 6 | 8 | 10 | |
| Immunogenicity <sup>i</sup> | | | X | X | X | X | X | | | | | X | | X | X |
| Biomarker storage sample | X | X | X | | X | | X | | | X | | | | X | X |
| CCI | | | | | | | | | | | | | | | |
| PK blood sample <sup>i</sup> | | | | X | X | X | X | X | X | X | X | X | X | X | X |
| CCI | | | | | | | | | | | | | | | |
| RNA | | | X | | | | | | | | | X | | X | |
| Study drug administered <sup>k</sup> | | | X | | X | X | X | X | | X | | | | | |
| Scales, Questionnaires, and | d Outcome N | leasures | | | | | | | | | | | | | |
| MIDAS | | | X | | | | X | | | | | X | | X | X |
| MSQ v2.1 | | | X | | X | X | X | X | | X | | X | | X | X |
| Non-migraine chronic pain assessment <sup>1</sup> | | | X | | | | X | | | | | X | | | X |
| PGI-S | | | X | | X | X | X | X | | X | | X | | X | X |
| PGI-I | | | | | X | X | X | X | | X | | X | | | X |
| C-SSRS/SHSF, SHFU <sup>m</sup> | X | X | X | | X | X | X | X | | X | | X | X | X | X |

Abbreviations: AE = adverse event; CGRP = Calcitonin-gene related peptide; C-SSRS = Columbia-Suicide Severity Rating Scale; ECG = electrocardiogram; ePRO = electronic patient reported outcomes; ET = early termination; FSH = follicle stimulating hormone; HDL = High-density lipoprotein; MIDAS = Migraine Disability Assessment test; MSQ (v2.1) = Migraine Specific Quality of Life Questionnaire; PGI-I = Patient Global Impression of Improvement; PGI-S = Patient Global Impression of Severity; PK = pharmacokinetics; RNA = ribonucleic acid; SHSF = Self-harm supplement form; SHFU = Self-harm follow-up form.

Note: Selected tests may be obtained in the event of a treatment-emergent hepatic abnormality and may be required in follow-up with patients in consultation with the Lilly, or its designee, clinical research physician. See Appendix 4 for more details regarding specific hepatic monitoring tests. If the patient has discontinued the trial and returns for hepatic follow-up, the site should use the 800 series as the visit designation.

#### Schedule of Activities, Protocol I5Q-MC-CGAH (footnotes)

- a The eligibility period of the prospective baseline assessment will last from 30 to 40 days. Investigators and patients may have up to an additional 5 days to schedule their Visit 3 appointment (beyond the 40 days); however, eligibility will be based on the 30-40 day period.
- b Visit is to include a review of any spontaneously reported adverse events and collection of blood samples for immunogenicity, PK, and CGRP plasma.
- c Visit 9 and Visit 11 are laboratory visits (for PK and CGRP plasma) only. Adverse events are not intended to be collected at these visits because patients may be going to a different location for laboratory assessments. However, any spontaneously reported AEs at these lab visits should be reported on the AE page.
- d A neurological exam will be conducted at screening, Month 3 and Month 6 of treatment, as well as at the final visit of the follow-up period or early termination visit in order to assess for any signs of pre-existing or treatment-emergent neurological abnormalities such as stroke or other cerebrovascular events.
- Electrocardiograms (ECGs) will be performed at Visit 1, Visit 3, Visit 12, and Visit 14 or early termination. Note: The Visit 3 ECG should be collected prior to blood draws and dosing. Patients must be supine for approximately 5 to 10 minutes before ECG collection and remain supine but awake during ECG collection.
- f Vital signs will include body temperature, blood pressure and pulse. Blood pressure and pulse will be measured in triplicate in the sitting position and should be measured prior to blood draws. Blood pressure will be assessed by utilizing a calibrated machine.
- g Chemistry samples collected at Visit 3, Visit 7, Visit 12, and Visit 14 or early termination must be fasting. Fasting is defined as no food or drink, except water, for at least 8 hours prior to testing.
- h In the event of a positive urine leukocyte esterase result, a repeat urine sample will be collected and shipped to the central laboratory.
- i A positive urine test must be followed by a serum pregnancy test for confirmation.
- Immunogenicity, CCl and PK sampling to be performed at the indicated visits and prior to dose administration if the visit is a dosing visit. Samples will be taken in the event of early termination. Immunogenicity samples also may be collected in the event of a systemic allergic/hypersensitivity reaction (see Section 8.4.3). The timing of samples will be recorded.
- k Patients will receive injections of placebo or LY2951742 after all other visit procedures are completed. Following the first dose at Visit 3, patients will be observed for at least 30 minutes in the office.
- 1 Questionnaire administered by clinician to assess other chronic pain conditions.
- m The C-SSRS and SHSF (and SHFU when applicable) will be completed at scheduled and unscheduled office visits.

# **Appendix 3.** Clinical Laboratory Tests

Hematology: Clinical Chemistry<sup>b</sup>: Hemoglobin Serum Concentrations of:

Hematocrit Sodium

Erythrocyte count (RBC) Potassium

Mean cell volume Total bilirubin

Mean cell hemoglobin concentration Direct bilirubin

Leukocytes (WBC) Alkaline phosphatase

Neutrophils, segmented Alanine aminotransferase (ALT) Lymphocytes Aspartate aminotransferase (AST) Monocytes Blood urea nitrogen (BUN)

Eosinophils Creatinine
Basophils Uric acid
Platelets Calcium

HbA<sub>1c</sub> Glucose (fasting)<sup>b</sup>

Albumin

Creatine kinase (CK)
Triglycerides
Total cholesterol<sup>b</sup>

 $HDL^b$ 

**Urinalysis**: Specific gravity

Urine culture<sup>a</sup>

рН

Insulin (fasting)<sup>b</sup> C-peptide (fasting)<sup>b</sup>

Protein Other CCI

Ketones PK Sample (LY2951742 serum concentration

Blood determination)
Urine leukocyte esterase<sup>a</sup> Immunogenicity
Microscopic analysis<sup>a</sup> Urine Drug Screen<sup>c</sup>

Pregnancy Test (females only)<sup>c</sup>
Serum pregnancy or FSH
Urine pregnancy test (local)

Stored Samples
Biomarker storage

RNA

Abbreviations: FSH = follicle-stimulating hormone; HDL = high density lipoprotein;

PK = pharmacokinetic; RBC = red blood cells; RNA = ribonucleic acid; WBC = white blood cells.

### **Clinical Laboratory Tests (footnotes)**

- <sup>a</sup> A positive urine leukocyte esterase result will require a follow-up sample with microscopic analysis and possibly a urine culture.
- Fasting laboratory samples will be collected as shown in the Schedule of Activities (Appendix 2). Fasting is defined as no food or drink, except water, for at least 8 hours prior to testing. All other samples may be collected on a nonfasting basis.
- <sup>c</sup> May be repeated during the study at the discretion of the investigator.

# Appendix 4. Hepatic Monitoring Tests for Treatment-Emergent Abnormality

Selected tests may be obtained in the event of a treatment-emergent hepatic abnormality and may be required in follow-up with patients in consultation with the Lilly, or its designee, clinical research physician.

### **Hepatic Monitoring Tests**

| Hepatic Hematologya | Haptoglobin <sup>a</sup> |
|--------------------------------|------------------------------------------|
| Hemoglobin | |
| Hematocrit | Hepatic Coagulationa |
| RBC | Prothrombin Time |
| WBC | Prothrombin Time, INR |
| Neutrophils, segmented | |
| Lymphocytes | Hepatic Serologies <sup>a,b</sup> |
| Monocytes | Hepatitis A antibody, total |
| Eosinophils | Hepatitis A antibody, IgM |
| Basophils | Hepatitis B surface antigen |
| Platelets | Hepatitis B surface antibody |
| | Hepatitis B Core antibody |
| Hepatic Chemistry <sup>a</sup> | Hepatitis C antibody |
| Total bilirubin | Hepatitis E antibody, IgG |
| Direct bilirubin | Hepatitis E antibody, IgM |
| Alkaline phosphatase | |
| ALT | Anti-nuclear antibodya |
| AST | Alkaline phosphatase isoenzymesa |
| GGT | Anti-Actin antibodya |
| CPK | Anti-smooth muscle antibody <sup>a</sup> |

Abbreviations: ALT = alanine aminotransferase; AST = aspirate aminotransferase; CPK = creatinine phosphokinase; GGT = gamma-glutamyl transferase; Ig = immunoglobulin; INR = international normalized ratio; RBC = red blood cells; WBC = white blood cells.

a Assayed by Lilly-designated or local laboratory.

b Reflex/confirmation dependent on regulatory requirements and/or testing availability.

# Appendix 5. Protocol Amendment I5Q-MC-CGAH(a) Summary: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients with Episodic Migraine – the EVOLVE-2 Study

### **Overview**

Protocol I5Q-MC-CGAH (CGAH) [A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients with Episodic Migraine – the EVOLVE-2 Study] has been amended. The new protocol is indicated by amendment (a) and will be used to conduct the study in place of any preceding version of the protocol.

The changes were required by 4 European Union Member States participating in the Voluntary Harmonisation Procedure. The key changes are as follows:

- Added the protocol amendment approval date (with updated trial alias) on every page of the protocol.
- Added language regarding the contents of each injection for the different treatment assignments in order to clarify how treatment is blinded (Section 4.1).
- Excluded patients with a prior lifetime history of stroke (Section 5.2, Exclusion [23]) to provide additional safeguards for patients who may be at risk for stroke.
- Added text to indicate that neurological examinations will be conducted to assess for possible cerebrovascular events, along with instructions for appropriate follow-up (Section 8.4.5, Safety Monitoring).
- Revised wording regarding procedures associated with emergency unblinding (Section 6.3) such that investigators no longer need to contact Lilly prior to emergency unblinding of a patient's treatment assignment.
- Added the list of allowed and disallowed concomitant treatments directly into Section 6.8 rather than referencing a separate document.
- Modified treatment discontinuation criteria (Section 7.1.1) to require (rather than recommend) discontinuation of treatment in the event of specific liver function test abnormalities, and added language to indicate the additional events requiring discontinuation from LY2951742 or placebo.
- Added information regarding the approximate number of countries, investigative sites, and patients planned for inclusion in Study CGAH (Section 9.1).



- Added clarification on the statistical model to be used for subgroup analyses (Section 9.7.2).
- Provided language clarifying the timing, and intent, of planned interim analyses (Section 9.8).
- Updated the Schedule of Activities and footnotes to reflect added neurological examinations.

### **Revised Protocol Sections**

#### Header

I5Q-MC-CGAH(a) Clinical Protocol

#### **Footer**

Approved: XX January 2016

#### **Title**

Protocol I5Q-MC-CGAH(a)

# 4. Study Design

### 4.1 Overview of Study Design

Patients randomized to the 120 mg dose of LY2951742 will receive an initial loading dose of 240 mg (2 injections of 120 mg each at Visit 3 only). To preserve blinding throughout the study, patients in all treatment groups will receive 2 injections of investigational product at each dosing visit (two placebo injections, two 120-mg LY2951742 injections, or one placebo injection and one 120-mg injection). At Visit 3, if available and where local regulations and Ethical Review Boards allow, patients will also watch a training video designed to address patient expectations with regard to participation in a placebo-controlled trial and the difference between medical treatment and research.

Patients will be given injections of investigational product during office visits (Figure CGAH.1). For all treatment groups, subcutaneous injections will be administered once monthly at the dosing visits. At Visit 3 (first dose), patients will be required to remain in the office for observation for 30 minutes post injection. Patients will continue to log in and complete the ePRO diary each day. Patients may continue to take their allowed acute migraine headache medication (with some limitations; see Section 6.8 concomitant medication study tool) during the treatment phase.

**Study Period IV**: During this 4-month phase, sites and patients will remain blinded to patients' treatment assignments. Patients will follow all study procedures during Study Period IV but will not receive LY2951742 or placebo. One month after Visit 12, if clinically warranted due to a worsening of symptoms, patients may start migraine prevention medications at the discretion of the investigator. The list of allowed preventive medications is provided in <u>Section 6.8 the concomitant medications study tool</u>. At Visit 14 (Month 10), patients will return to the site for their last study visit and discharge from the study.

### 5.2 Exclusion Criteria

#### **Medical Conditions**

[23] Have ECGs showing abnormalities compatible with acute cardiovascular events and/or serious cardiovascular risk, including but not limited to a corrected QT (QTcB [Bazett's]) interval > 470 msec for women and >450 for men, or have had myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, stroke, or deep vein thrombosis/pulmonary embolism within 6 months of screening, or have planned cardiovascular surgery or percutaneous coronary angioplasty, or patients with a lifetime history of stroke.

### 5.3 Screen Failures

Individuals who do not meet the criteria for participation in this study (screen failure) may be considered for rescreen once, with approval from Lilly Medical for only the criteria shown below. The interval between screening and rescreening must be at least 45 days or longer if required for the specified timeframes in the inclusion/exclusion criteria or concomitant medications requirements study tool. If rescreening is performed, the individual must sign a new ICF and will be assigned a new identification number.

# 6.3 Blinding

In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a patient's treatment assignment is warranted. Patient safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the Lilly CRP/CRS prior to unblinding a patient's treatment assignment. If an emergency unblinding occurs, a patient's treatment assignment is unblinded, Lilly must be notified as soon as possible immediately.

# 6.8 Concomitant Therapy

Table CGAH.3 contains a list of medications that are, and are not, allowed in this study. Note that acute treatment of migraine headache is allowed throughout the study but with some limitations. Treatments used for the prevention of migraine are not allowed at any time during Study Periods I through III.

# <u>Table CGAH.3.</u> <u>Treatments Allowed and Treatments Not Allowed as Concomitant</u> Therapy

# Medications allowed for the ACUTE treatment of migraine headaches or other pain or injury:

Acetaminophen (paracetamol), NSAIDs; Triptans; Ergotamine and derivatives; Isometheptene mucate, dichloralphenazone and acetaminophen combination (Midrin); or combinations thereof.

The following medications are allowed with restrictions:

- 3. Opioid and barbiturates no more than 3 days/month (SP II, III and IV).
- 4. Single dose of injectable steroids allowed only once during the study, in an emergency setting (SP III and IV).

### Medications, Procedures or Devices not allowed for any reason/indication:

Acetazolamide

Acupuncture

Anticonvulsants/Antiepileptics

Antipsychotics

Beta-blockers

Botulinum toxin applied to head/neck area

Cannabis / Cannabinoids

Chiropractic procedures, physiotherapy, TENS or other electric devices on head and neck

Corticosteroids for oral use

Flunarizine

Herbals with anti-inflammatory effect (feverfew, willow bark, petasites/butterbur), herbals with sympathomimetic effect (ma huang, ephedra, bitter orange, synephrine) and herbals with catecholamine transmitter reuptake inhibition (St John's Wort)

Monoamine oxidase inhibitors (MAOIs)

**Memantine** 

Serotonin 5HT2a/2c antagonists, ege.g.: trazodone, nefazodone

Stimulants (prescription strength), ege.g.: methylphenidate, dextroamphetamine, mixed amphetamine salts

**Tizanidine** 

Therapeutic antibodies, ege.g.: adalimumab, infliximab, trastuzumab, bevacizumab, etanercept, etc.

Tricyclic antidepressants (TCAs)

Triptans for prophylaxis of menstrual related migraine

Venlafaxine

Verapamil

# Restricted medication during SP II-III: Use of the following medications for indications other than migraine prevention is allowed providing the dose is stable 2 months prior to Visit 2 and is expected to remain stable during Visit 2 through-V12.

**ACE** inhibitors

Angiotensin receptor blockers (ARBs)

Benzodiazepines

Bupropion

Calcium-channel blockers (except verapamil and flunarizine)

Clonidine

Guanfacine

**Mirtazapine** 

SSRIs/NRIs/SNRIs (other than venlafaxine)

Use of electric devices (i.e. TENS), physiotherapy, chiropractic procedures on low back and extremities

# Restricted medication during SP II-III: Use of the following medications for indications other than migraine prevention is allowed:

Beta-blockers, ophthalmic

Cyclandelate

Cyproheptadine

Melatonin

### SP IV (After Visit 12)

One month after Visit 12, if clinically warranted due to a worsening of symptoms, patients may start migraine prevention medications at the discretion of the investigator with the exception of antipsychotics, cannabis and cannabinoids, MAOIs, memantine, serotonin 5HT2a/2c antagonists, and stimulants, which remain excluded.

The list of medications allowed or not allowed for the acute treatment of migraine, as well as those prohibited for the prevention of migraine, is provided in the concomitant medication list in the concomitant medications study tool, along with all concomitant therapies allowed or not allowed during the study. Note that there are some limitations regarding concomitant medications for the acute treatment of migraines during the study. Any changes in the list of allowed/not allowed medications will be communicated to investigators and will not constitute a protocol amendment.

# 7. Discontinuation Criteria

# 7.1 Discontinuation from Study Treatment

# 7.1.1. Permanent Discontinuation from Study Treatment

Discontinuation of the investigational product is required in cases of pregnancy.

Discontinuation of the investigational product for abnormal liver tests <u>is required</u>should be considered by the investigator when a patient meets one of the following conditions <u>and the event is at least possibly related to study drugafter consultation with the Lilly designated medical monitor:</u>

- ALT or aspartate aminotransferase (AST) >8X ULN
- ALT or AST >5X ULN for more than 2 weeks
- ALT or AST >3X ULN and TBL >2X ULN or prothrombin time >1.5X ULN

- ALT or AST >3X ULN with the appearance of fatigue, nausea, vomiting, right upper-quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)
- ALP >3X ULN
- ALP >2.5X ULN and TBL >2X ULN
- ALP >2.5X ULN with the appearance of fatigue, nausea, vomiting, right quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%)

Discontinuation of investigational product also is required in the following cases, if the event is at least possibly related to study drug:

- Serious allergic reaction to study drug
- <u>Serious injection-site reaction</u>
- Serious event of suicidality or depression
- Serious cerebrovascular event.

# 8. Study Assessments and Procedures

# 8.4 Safety Assessments

# 8.4.5 Safety Monitoring

Neurological examinations will be conducted at screening, Month 3 and Month 6 of treatment, as well as at the final visit of the follow-up period or early termination visit in order to assess for any signs of pre-existing or treatment-emergent neurological abnormalities such as stroke or other cerebrovascular events. If a study patient experiences signs of a cerebrovascular event, appropriate follow-up and clinical management should be conducted by the investigator, and the Lilly CRP/CRS should be consulted regarding collection of further clinical information and follow-up testing.

# 9. Statistical Considerations and Data Analysis

# 9.1 Determination of Sample Size

Approximately 100 sites in 11 countries are planned for inclusion in Study CGAH, with an average of approximately 8 patients to be randomized at each investigative site. The final number of sites, countries, and patients per site may vary depending on sites' enrollment rates.

### 9.2 General Statistical Considerations

The primary analysis will be performed using a restricted maximum likelihood-based mixed models repeated measures (MMRM) technique with prespecified model terms (Section 9.4.1).

Any change to the data analysis methods described in the protocol will require an amendment ONLY if it changes a principal feature of the protocol. Any other change to the data analysis methods described in the protocol, and the justification for making the change, will be described in the clinical study report or SAP. Changes may only be made in the SAP prior to unblinding. Additional exploratory analyses of the data will be conducted as deemed appropriate.

# 9.4 Primary and Secondary Analyses

# 9.4.2. Key Secondary Analyses





There will be no adjustments for multiplicity for analyses of other endpoints. If the multiple testing approach for key secondary measures only needs to be changed, the updated approach will be provided in the SAP, and it should not lead to modification of this protocol.

# 9.7.2 Subgroup Analyses

Subgroup analyses will be performed for the primary efficacy measure (change from baseline in the number of migraine headache days) <u>separately for each of the subgroup populations listed in Table CGAH.4.</u> Subgroup analyses will be conducted only for the ITT patients in Study Period III.

Each of tThe subgroup analyses for the primary measure of change from baseline in the number of migraine headache days will be conducted using MMRM. The same MMRM model described in Section 9.4.1 will be used, with terms of subgroup, subgroup-by-treatment, subgroup-by-month, and subgroup-by-treatment-by-month interactions added as additional covariates.

### Table CGAH.34. Definition of Subgroup Variables

### 9.8 Interim Analyses

Two interim analyses are anticipated for this study. The first possible interim analysis will occur during Study Period III (double-blind treatment) and could result in stopping the trial for safety or futility. Details will be documented in the Statistical Analysis Center SAP and the DMC Charter. A DMC will be convened to assess safety and futility analyses. This analysis is planned to occur when approximately 330 (40% of the total sample size) randomized patients have had the chance to complete at least 3 months of the treatment period. The interim analysis will be conducted by an independent data monitoring committee (DMC) with members external to Lilly. The data from the interim analysis will be used to evaluate whether to stop or modify the study for futility and/or safety issues. Stopping rules for futility at this interim analysis will be based on the conditional power of comparing LY2951742 to placebo. Specifically, conditional power represents the probability that the ongoing trial will result in a statistically significant difference between LY2951742 and placebo at end of the trial, based on the data available at the time of the interim analysis. Rules for stopping the study are detailed in the Statistical Analysis Center SAP and the DMC Charter. Only the DMC is authorized to evaluate unblinded interim efficacy and safety analyses. Study sites will receive information about interim results ONLY if they need to know for the safety of their patients. There is no inflation of type 1 error due to the conduct of a futility analysis (Snapinn et al. 2006), so no adjustment to the nominal significance level will be made for the primary analysis as a result of a futility assessment.



# **Appendix 2** Schedule of Activities

Schedule of Activities, Protocol I5Q-MC-CGAH

| Study Period (SP) | SP I-<br>Screening | SP II-<br>Prospective<br>Baseline | | SP III - Treatment | | | | | | | | | | SP IV – Follow-u | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (Target) Interval (days)<br>since previous visit | | | 30-45 | 14 | 16 | 30 | 30 | 30 | 15 | 15 | 15 | 15 | 60 | 60 | |
| Allowable range (days)<br>between visits | 3-45 | 30-40 <sup>a</sup> | | | | | | | | | | | | | |
| Interval allowance (days) | | | | +/- 1 | +/- 3 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 2 | +/- 5 | +/- 5 | ET |
| Visit | 1 | 2 | 3 | 4b | 5 | 6 | 7 | 8 | 9° | 10 | 11° | 12 | 13 | 14 | |
| Month | | | 0 | 0.5 | 1 | 2 | 3 | 4 | 4.5 | 5 | 5.5 | 6 | 8 | 10 | |
| Assessments and Procedur | es | | | | | | | | | | | | | | |
| Physical examination <sup>d</sup> | X | | | | | | | | | | | | | | |
| Neurological<br>examinationd | <u>X</u> | | | | | | <u>X</u> | | | | | <u>X</u> | | <u>X</u> | <u>X</u> |

### Schedule of Activities, Protocol I5Q-MC-CGAH (footnotes)

d Physical examinations at screening must include a neurological exam. A neurological exam will be conducted at screening. Month 3 and Month 6 of treatment, as well as at the final visit of the follow-up period or early termination visit in order to assess for any signs of pre-existing or treatment-emergent neurological abnormalities such as stroke or other cerebrovascular events.

Leo Document ID = 0141c58f-0217-46f5-9eb1-151a7b7010e3

Approver: PPD

Approval Date & Time: 22-Jan-2016 16:59:38 GMT

Signature meaning: Approved

Approver: PPD

Approval Date & Time: 22-Jan-2016 20:45:52 GMT

Signature meaning: Approved